

## STATISTICAL ANALYSIS PLAN VERSION: 2.0

# A RANDOMIZED, DOUBLE-MASKED, ACTIVE-CONTROLLED PHASE 2/3 STUDY OF THE EFFICACY AND SAFETY OF HIGH-DOSE AFLIBERCEPT IN PATIENTS WITH DIABETIC MACULAR EDEMA

High-dose aflibercept

| - | • |
|---------------------------|--------------------------------------|
| Study Name | PHOTON |
| Protocol Number: | VGFTe-HD-DME-1934 |
| Clinical Phase: | 2/3 |
| Sponsor: | Regeneron Pharmaceuticals, Inc. |
| Study Biostatisticians: | |
| Project Biostatisticians: | |
| Clinical Trial Manager: | |
| Study Medical Director: | |
| Version/Date: | Original (Version 1.0) / 05 JUL 2022 |
| | Amendment Version 2.0 / 19 AUG 2022 |

CONFIDENTIAL Document's type Standard

**Compound:** 

 Document Reference BDM-STD-STA4-2.2

Effective Date March 1, 2015

Statistical Analysis Plan Date: 19 AUGUST 2022

Protocol: VGFTe-HD-DME-1934

The approval signatures below indicate that these individuals have reviewed the Statistical Analysis Plan (SAP) and agreed on the planned analysis defined in this document for reporting.

| See appended electronic signature page |
|----------------------------------------|
| Study Biostatistician |
| See appended electronic signature page |
| Study Pharmacokinetics |
| See appended electronic signature page |
| Study Bioanalytical Sciences |
| See appended electronic signature page |
| Study Medical Director |
| See appended electronic signature page |
| Project Biostatistician |
| See appended electronic signature page |
| Head of BDM or designee |

### Protocol: VGFTe-HD-DME-1934 Date: 19 AUGUST 2022

## **TABLE OF CONTENTS**

| LIST OF | F ABBREVIATIONS AND DEFINITION OF TERMS | 7 |
|---|---|---|
| 1. | OVERVIEW | 10 |
| 1.1. | Background/Rationale | 10 |
| 1.2. | Study Objectives | 11 |
| 1.2.1. | Primary Objectives | 11 |
| 1.2.2. | Secondary Objectives | 11 |
| 1.2.3. | Exploratory Objectives | 11 |
| 1.2.4. | Modifications from the Statistical Section in the Final Protocol | 11 |
| 1.2.5. | Revision History for SAP Amendments | 12 |
| 2. | INVESTIGATION PLAN | 13 |
| 2.1. | Study Design and Randomization | 13 |
| 2.2. | Sample Size and Power Considerations | 16 |
| 3. | ANALYSIS POPULATIONS | 17 |
| 3.1. | The Full Analysis Set (FAS) | 17 |
| 3.2. | The Per Protocol Set (PPS) | 17 |
| 3.3. | The Safety Analysis Set (SAF) | 17 |
| 3.4. | Pharmacokinetic Analysis Sets | 17 |
| 3.5. | Immunogenicity Analysis Sets | 18 |
| 4. | ANALYSIS VARIABLES | 19 |
| 4.1. | Demographic and Baseline Characteristics | 19 |
| 4.2. | Medical History | 20 |
| 4.3. | Pre-Treatment / Concomitant Medication | 20 |
| 4.4. | Exposure, Compliance, Additional Treatment to Study Treatment | 20 |
| 4.5. | Efficacy Variable | 21 |
| 4.5.1. | Primary Efficacy Variable (s) | 21 |
| 4.5.2. | Key Secondary Efficacy Variable(s) | 21 |
| 4.5.3. | Additional Secondary Efficacy Variable(s) | 21 |
| 4.5.4. | Exploratory Efficacy Variable(s) | 21 |
| 4.6. | Safety Variables | 23 |
| 4.6.1. | Adverse Events and Serious Adverse Events | 23 |
| 4.6.2. | Laboratory Safety Variables | 23 |

| 23 |
|----|
| 23 |
| 24 |
| 24 |
| 24 |
| 24 |
| 25 |
| 25 |
| 25 |
| 25 |
| 25 |
| 26 |
| 26 |
| 26 |
| 28 |
| 30 |
| 30 |
| 31 |
| 32 |
| 32 |
| 33 |
| 33 |
| 33 |
| 34 |
| 34 |
| 35 |
| 36 |
| 36 |
| 37 |
| 38 |
| 38 |
| 38 |

| 5.7.5. | Analysis of Other Ocular Safety Variables | 39 |
|---|---|---|
| 5.7.6. | Surgeries | 39 |
| 5.8. | Analysis of Pharmacokinetic Data | 39 |
| 5.8.1. | Analysis of Drug Concentration Data | 39 |
| 5.8.2. | Pharmacokinetics/Pharmacodynamics Analyses | 40 |
| 5.9. | Analysis of Immunogenicity Data | 40 |
| 6. | DATA CONVENTIONS | 42 |
| 6.1. | Definition of Baseline | 42 |
| 6.2. | Visit Windows | 42 |
| 6.3. | Unscheduled Assessments | 42 |
| 6.4. | Handling of Patients who Discontinue | 42 |
| 6.5. | Data Handling Convention for Missing Data | 42 |
| 7. | INTERIM ANALYSIS | 44 |
| 8. | SOFTWARE | 45 |
| 9. | REFERENCES | 46 |
| 10. | APPENDIX | 47 |
| 10.1. | Summary of Statistical Analyses | 47 |
| 10.2. | Schedule of Time and Events | 53 |
| 10.2.1. | Schedule of Time and Events (Main study) | 53 |
| 10.2.2. | Schedule of Time and Events (Dense PK substudy) | 58 |
| 10.3. | NEI-VFQ-25 Sub-scale Scores and Total Score | 59 |
| 10.4. | Detailed Definitions of Special AE Categories and Medical History<br>Subgroups | 60 |
| 10.4.1. | Medical history and AE grouping of hypertension | 60 |
| 10.4.2. | AE grouping of intraocular inflammation | 62 |
| 10.4.3. | AE grouping of nasal mucosal events | 63 |
| 10.4.4. | Medical history of renal impairment | 63 |
| 10.4.5. | Medical history of hepatic impairment | 64 |
| 10.4.6. | Medical history of cerebrovascular disease | 75 |
| 10.4.7. | Medical history of ischemic heart disease | 82 |
| 10.5. | Criteria for Potentially Clinically Significant Values (PCSV) | 84 |
| 10.6. | Process to Derive Week 48 Data Cut-off | 86 |
| 10.6.1. | Visit Independent Data | 86 |

| _ | Analysis Plan | rotocol: VGFTe-HD-DME-1934<br>Date: 19 AUGUST 2022 |
|---|---|---|
| 10.6.2. | Study Medication Data | 87 |
| 10.6.3. | Visit Dependent Data | 87 |
| 10.7. | Process to Derive Week 60 Data Cut-off | 88 |
| 10.8. | SAS Procedures | 88 |
| 10.8.1. | MMRM | 88 |
| 10.8.2. | ANCOVA | 88 |
| 10.8.3. | Multiple Imputation | 88 |
| 10.8.4. | Tipping Point Analysis | 89 |
| 10.9. | Additional Secondary Efficacy Variables and Analys | es91 |
| 10.9.1. | Analysis Populations | 91 |
| 10.9.1.1. | Full Analysis Set (FAS) | 91 |
| 10.9.1.2. | Modified Full Analysis Set (mFAS) | 91 |
| 10.9.2. | Additional Secondary Efficacy Variable(s) | 91 |
| 10.9.3. | Additional Secondary Efficacy Analyses | 92 |
| | LIST OF TABLES | |
| Table 1: S | trategies for occurrence of intercurrent events (ICE) | 27 |
| Table 2: T | he Testing Order of Hierarchical Testing Procedure in | G-SAP and EP-SAP35 |
| Table 3: R | ecoding of NEI-VFQ 25 items | 59 |
| Table 4: S | ub-scales of the NEI-VFQ 25 score | 60 |
| Table 5: C | riteria for Potentially Clinically Significant Values | 84 |
| Table 6: A | Additional Secondary Efficacy Analyses – Alternative | Tipping Point Analyses93 |
| | LIST OF FIGURES | |
| Figure 1: S | Study Flow Diagram | 14 |

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

2q8 2 mg aflibercept every 8 weeks

AAS ADA analysis set
ADA Anti-drug antibody
AE Adverse event

ALT Alanine aminotransferase ANCOVA Analysis of covariance

APTC Anti-Platelet Trialists' Collaboration

AST Aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

BCVA Best corrected visual acuity

BMI Body mass index
BP Blood pressure

BRVO Branch retinal vein occlusion

BUN Blood urea nitrogen
CI Confidence interval

CMH Cochran Mantel Haenszel
CPK Creatine phosphokinase

CRF Case report form

CRT Central retinal thickness

CRVO Central retinal vein occlusion

CSME Clinically Significant Macular Edema

DME Diabetic macular edema
DPKS Dense PK analysis set
DR Diabetic retinopathy

DRM Dose Regimen Modification

DRSS Diabetic Retinopathy Severity Scale

ECG Electrocardiogram

EMA European Medicines Agency

EP-SAP Statistical analysis plan for EMA and PMDA

EOS End of study

ETDRS Early Treatment Diabetic Retinopathy Study

FA Fluorescein angiography

FAS Full analysis set

G-SAP Global statistical analysis plan


Regeneron Pharmaceuticals, Inc.

Statistical Analysis Plan

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

HbA1c Hemoglobin A1c

HD High-dose

HDq12 High-dose aflibercept every 12 weeks HDq16 High-dose aflibercept every 16 weeks

HDL High-density lipoprotein ICF Informed consent form

ICE Intercurrent event

ICH International Council for Harmonisation

IOP Intraocular pressure IRF Intraretinal fluid

IVT Intravitreal

IWRS Interactive web response system LOCF Last observation carry forward

LDH Lactate dehydrogenase
LDL Low-density lipoprotein

LS Least square

MAR Missing at random
MI Multiple imputation

MCMC Markov Chain Monte Carlo

mCNV Myopic choroidal neovascularization

MedDRA Medical Dictionary for Regulatory Activities

(MedDRA) HLT High Level Term

MMRM Mixed-model repeated measures

NAb Neutralizing antibody NAbAS NAb analysis set

nAMD Neovascular "wet" age-related macular degeneration

NEI-VFQ-25 National Eye Institute Visual Functioning Questionnaire-25

OC Observed case

OCT Optical coherence tomography

PCSV Potentially clinically significant value

PK Pharmacokinetic PKAS PK analysis set

PMDA Pharmaceuticals and Medical Devices Agency

PPS Per protocol set
PT Preferred term
RBC Red blood cell

Protocol: VGFTe-HD-DME-1934 Statistical Analysis Plan Date: 19 AUGUST 2022

SAE Serious adverse event SAF Safety analysis set SAP Statistical analysis plan SAS Statistical Analysis System

SD Standard deviation

**SD-OCT** Spectral domain optical coherence tomography

Standard international SI SOC System organ class SRF Subretinal fluid

TEAE Treatment-emergent adverse event

**UPCR** Urine protein:creatinine ratio

VA Visual acuity

**VEGF** Vascular endothelial growth factor

WBC White blood cell

WHODD World Health Organization Drug Dictionary

#### 1. **OVERVIEW**

The purpose of the statistical analysis plan (SAP) is to ensure the credibility of the study results by pre-specifying the statistical approaches for the analysis of study data prior to database lock. The SAP is intended to be a comprehensive and detailed description of the strategy and statistical methods to be used in the analysis of data for the phase 2/3 PHOTON, VGFTe-HD-DME-1934, study of high-dose (HD) aflibercept in patients with Diabetic Macular Edema (DME). This SAP is based on Protocol Amendment 4 dated April 28, 2022.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

## 1.1. Background/Rationale

Diabetic retinopathy (DR) is the most common microvascular complication of diabetes. DME, a manifestation of diabetic retinopathy, is the primary cause of vision loss and blindness in patients with diabetes and the most frequent cause of blindness in young and middle-aged adults. If left untreated, approximately half of patients with DME will lose 2 or more lines of visual acuity (VA) within 2 years.

Treatment options for DME include laser photocoagulation and pharmacologic interventions, specifically vascular endothelial growth factor (VEGF) inhibitors and steroids. Surgery is also performed in some cases as a fall-back therapeutic option, particularly for those refractory to treatment or with vitreomacular traction.

However, anti-VEGF compounds have become the standard of care for the treatment of DME. This approach is highly attractive as it directly targets VEGF, one of the main mediators of DR and DME. Vascular endothelial growth factor is a protein growth factor that both stimulates angiogenesis and increases vascular permeability, playing a key role in the pathophysiology of DME. Hypoxia and other metabolic factors trigger VEGF release. VEGF induces vascular leakage and neovascularization. While neovascularization is the most severe manifestation of DR, vascular leakage leading to macular edema is an important cause of reduced visual acuity.

EYLEA (also known as intravitreal aflibercept injection) is a VEGF antagonist currently approved in over 100 countries for the treatment of DME at a dosage level of 2 mg (administered at a concentration of 40 mg/mL injected intravitreally [IVT]). EYLEA is currently approved in at least 100 countries for additional indications that include neovascular age-related macular degeneration (nAMD), macular edema following central retinal vein occlusion (CRVO) and branch retinal vein occlusion (BRVO), and in 99 countries for the treatment of myopic choroidal neovascularization (mCNV). EYLEA is also approved in the United States for the treatment of diabetic retinopathy.

Despite available treatments, there remains an unmet medical need for the development of therapies with the potential to improve important clinical outcomes. This unmet need includes decreasing the treatment burden via a reduction in the required frequency of intravitreal injections, improving visual and anatomic outcomes over currently available standards of care, and slowing or even reversing the underlying pathophysiology of the disease itself, specifically retinal ischemia.

Increasing the drug product concentration of aflibercept allows a greater amount of drug to be delivered IVT and thus has the potential to increase aflibercept's pharmacological duration of action, and thereby provide additional benefit to patients with DME. The resulting extension of

treatment intervals to every 12 weeks or 16 weeks, early after the initiation of treatment, would reduce the number of injections in the first treatment year. A potential decrease in injection-related treatment burden and safety events could be a significant contribution to patient care and healthcare services.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

This Phase 2/3 study (hereafter referred to as PHOTON) is designed as a randomized, double-masked, active-controlled non-inferiority study to evaluate the safety and efficacy of a HD aflibercept with the intent of extending the dosing interval, with at least similar functional and potentially improved anatomic outcomes compared to the active control arm of 2 mg aflibercept (EYLEA). The PHOTON study will investigate HD aflibercept dosed every 12 weeks (HDq12) or 16 weeks (HDq16) after 3 initial monthly injections vs. 2 mg aflibercept dosed every 8 weeks (2q8) after 5 initial monthly injections in patients diagnosed with DME.

#### 1.2. Study Objectives

#### 1.2.1. Primary Objectives

The primary objective of the study is to determine if treatment with HD aflibercept at intervals of 12 or 16 weeks provides noninferior best corrected visual acuity (BCVA) compared to 2 mg aflibercept dosed every 8 weeks.

#### 1.2.2. Secondary Objectives

The secondary objectives of the study are as follows:

- To determine the effect of HD vs. 2 mg aflibercept on anatomic and other visual measures of response
- To evaluate the safety, immunogenicity, and pharmacokinetics (PK) of aflibercept.

#### 1.2.3. Exploratory Objectives

The exploratory objectives of the study are as follows:

- To determine the effect of HD vs. 2 mg aflibercept on additional anatomic measures of response
- To study molecular drivers of DME or related diseases, the mechanism of action of aflibercept, and the VEGF pathway

#### 1.2.4. Modifications from the Statistical Section in the Final Protocol

Additional secondary efficacy endpoints and their analyses are added to this SAP for submission to the US FDA (based on the G-SAP that constitutes the primary analysis for the study). See Appendix 10.9 for details.

## 1.2.5. Revision History for SAP Amendments

| Version | Date | Version history |
|---|---|---|
| 1.0 | 05 July 2022 | Initial version |
| 2.0 | 19 August 2022 | Additional secondary efficacy variables and their analyses are added to the Appendix 10.9 of the SAP |

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

#### 2. INVESTIGATION PLAN

## 2.1. Study Design and Randomization

This phase 2/3, multi-center, randomized, double-masked study in patients with DME involving the center of the macula will investigate the efficacy and safety of HD aflibercept versus 2 mg aflibercept.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

The study consists of a screening/baseline period, a treatment period, and an end of study (EOS) visit at week 96. A total of approximately 640 eligible patients will be randomized into 3 treatment groups in a 1:2:1 ratio as follows (Figure 1):

- 1. 2q8: 2 mg aflibercept every 8 weeks, following 5 initial monthly doses (n=160),
- 2. HDq12: HD aflibercept every 12 weeks, following 3 initial monthly doses (n=320),
- 3. HDq16: HD aflibercept every 16 weeks following 3 initial monthly doses (n=160).

Randomization of patients will be stratified based on

- baseline central retinal thickness (CRT) (<400 μm, ≥400 μm),
- prior DME treatment (yes, no), and
- geographical region (Japan, Rest of world).

Sham injections will be given at all visits when an active injection is not planned. All patients will be followed every 4 weeks through week 96.

The primary analysis will take place once all patients have completed week 48 (or prematurely discontinued), with additional analyses after all patients have completed week 60, and after all patients have completed the study at week 96.

Approximately 24 patients will be included in a dense PK substudy (n=8 per group, with half Japanese and half non-Japanese per group). For details refer to Appendix 10.2.2.

In all patients, blood samples for measurement of drug concentrations (PK) and anti-drug antibody (ADA) will be obtained prior to the first treatment and at prespecified time points throughout the course of the study (see Schedule of Events in Appendix 10.2). In addition, a DNA sample will be collected from those who sign the informed consent form (ICF) for the optional genomic substudy.

Dosing schedules appear in Figure 2 and are described below.

Protocol: VGFTe-HD-DME-1934 Date: 19 AUGUST 2022

Figure 1: Study Flow Diagram



\*Treatment Naïve and Previously Treated

Figure 2: Dosing Schedule

**PHOTON:** Dosing Schedule

| 2q8 | Х | х | х | х | х | 0 | х | 0 | х | 0 | х | 0 | Х |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| HDq12 | Х | Х | Х | 0 | 0^ | X^ | 0 | 0 | χa | 0 | 0 | Хa | 0 |
| HDq16 | х | Х | Х | 0 | o* | o* | Х* | 0 | 0 | 0 | Хa | 0 | 0 |
| ive injection | Oose Regime<br>Q12 group:<br>HDq16 grou<br>For patients<br>osing interv | If criteria a<br>up: If criteri<br>on a dosin | are met, pa<br>a are met<br>g interval | atients will<br>at week 16<br>of q12 or q | or 20, pat | ient will co | | | | | | | |
| ive injection | Q12 group:<br>HDq16 grou<br>For patients | If criteria a<br>up: If criteri<br>on a dosin | are met, pa<br>a are met<br>g interval | atients will<br>at week 16<br>of q12 or q | or 20, pat | ient will co<br>DRM crite | ia will be | assessed | at dosing v | | | | t the ne |
| ive injection | Q12 group:<br>HDq16 grou<br>For patients<br>osing interv | If criteria a<br>up: If criteri<br>on a dosin<br>val will be r | are met, pa<br>a are met<br>g interval<br>educed by | atients will<br>at week 16<br>of q12 or q<br>4 weeks. | or 20, pat<br>16 weeks, | ient will co<br>DRM crite | ia will be | assessed | at dosing v | isits and if | DRM crite | eria are me | |
| ive injection<br>im injections | Q12 group:<br>HDq16 grou<br>For patients<br>Josing interv | If criteria a<br>up: If criteri<br>on a dosin<br>val will be r<br>wk 56 | are met, pa<br>a are met<br>g interval<br>educed by | at week 16<br>of q12 or q<br>4 weeks. | or 20, pat<br>16 weeks,<br>Wk 68 | ient will co<br>DRM crite | ia will be | assessed | at dosing v | isits and if | DRM crite | eria are me | t the ne |

Note: Figure does not reflect all dosing options, once a patient is shortened or extended

#### **Dose Regimen Modifications/Rescue Regimen**

For masking purposes, assessments for dose regimen modifications (DRMs) will be performed in all patients at all visits (through the interactive web response system [IWRS]) beginning at week 16. Based on these assessments, patients in the HD groups may have their treatment intervals shortened (year 1 and year 2) or extended (year 2). The minimum interval between injections will be 8 weeks which is considered a rescue regimen for patients randomized to HD aflibercept and unable to tolerate a dosing interval greater than every 8 weeks. Patients in the aflibercept 2 mg group will remain on fixed q8 dosing throughout the study (ie, will not have modifications of their treatment intervals regardless of the outcomes of the DRM assessments)

#### Year 1: Baseline to Week 52

Beginning at week 16, patients in the HD groups will have the dosing interval shortened (at the visits described below) if BOTH of the following criteria are met:

1. > 10 letter loss in BCVA from week 12 in association with persistent or worsening DME AND

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

2. >50 μm increase in CRT from week 12

(It should be noted that the change in CRT for these criteria will be assessed at the site.)

If a patient in the HDq12 group or the HDq16 group meets both criteria at week 16 or week 20, the patient will be dosed with 8 mg aflibercept at that visit and will continue on a rescue regimen (aflibercept 8 mg, every 8 weeks). If a patient in the HDq16 group who has not met the criteria at week 16 or 20 meets both criteria at week 24, the patient will be dosed with 8 mg aflibercept at that visit and will continue on q12 week dosing.

For patients whose interval was not shortened to q8 dosing at or before week 24, the interval will be shortened if the DRM criteria are met at a subsequent dosing visit. Patients in the HDq12 group who meet the criteria will receive the planned dose at that visit and will then continue on a rescue regimen (aflibercept 8 mg, every 8 weeks). Patients in the HDq16 group who meet these criteria will receive the planned dose at that visit and will then continue to be dosed every 12 weeks if they were on a 16-week interval, or switch to the rescue regimen (aflibercept 8mg, every 8 weeks) if they were previously shortened to a 12-week interval. Therefore, a patient randomized to HDq16 whose injection interval has been shortened to q12 will have their injection interval further shortened to q8 if these criteria are met at any subsequent dosing visit.

#### Year 2: Week 52 to Week 96 (End of Study)

From week 52 through the end of study (year 2), all patients in the HD groups will continue to have the interval shortened in 4-week intervals if the DRM criteria for shortening are met at dosing visits using the DRM criteria described above for year 1. As in year 1, the minimum dosing interval for patients in all treatment groups is every 8 weeks.

In addition to shortening of the interval, all patients in the HD groups (including patients whose interval was shortened during year 1) may be eligible for interval extension (by 4-week increments), if BOTH the following criteria are met at dosing visits in year 2:

- 1. <5 letter loss in BCVA from week 12 AND
- 2. CRT <300 μm on Spectral domain optical coherence tomography (SD-OCT) (or <320 μm on Spectralis SD-OCT)

For patients who do not meet the criteria for shortening or extension of the interval, the dosing interval will be maintained.

As in year 1, all patients in all treatment groups (including the 2q8 group) will be evaluated against both DRM criteria at all visits through the IWRS for masking purposes. However, changes to dosing schedule will only be implemented as described above for those patients randomized to HDq12 or HDq16 treatment groups. No changes to the dosing schedule will be made to the 2q8 treatment group at any time.


## 2.2. Sample Size and Power Considerations

The sample size calculation is based on the primary endpoint, the change from baseline in BCVA at week 48 in 2 pairwise comparisons: (1) HDq12 vs. 2q8; (2) HDq16 vs. 2q8. The non-inferiority margin is defined to be 4 letters.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

Under the original testing strategy (prior to Amendment 4), assuming a standard deviation of 9.07 letters for each treatment group (Brown, 2015), a sample size of 129 patients per group will provide 90% power using a two-sample t-test to demonstrate non-inferiority with one-sided alpha=0.0125 (=0.025/2) for each comparison. The overall family-wise type I error rate of 0.025 (one-sided) will be preserved. Allowing for a dropout rate of 19%, 160 patients per group will be required to provide 90% power for each pairwise comparison. However, the sample size in the HDq12 group has been doubled to meet regulatory requirements for the safety database. This results in a total of 640 patients for 3 groups (160, 160, and 320 patients for groups 2q8, HDq16, and HDq12, respectively). Therefore, with these sample sizes, the power for the pairwise comparisons will be: 90% for HDq16 vs. 2q8, and approximately 97% for HDq12 vs. 2q8. The power to reject each of the primary hypotheses with the proposed multiple testing procedure will be at least as high. Sample size/power calculations were performed using East 6 software.

However, under the current hierarchical testing procedure, using the same assumptions as indicated above, a total sample size of 640 patients for 3 groups provides 98% power for the comparison of HDq12 vs. 2q8, and subsequently 92% power for the comparison of HDq16 vs. 2q8, for the primary endpoint assessing non-inferiority, with a 1-sided t-test at significance level of 0.025.

#### 3. ANALYSIS POPULATIONS

In accordance with guidance from the International Conference of Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) guideline ICH E9 Statistical Principles for Clinical Trials (ICH, 1998), the following population of analysis will be used for all statistical analysis:

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

## 3.1. The Full Analysis Set (FAS)

The full analysis set (FAS) includes all randomized patients who received at least 1 dose of study medication; it is based on the treatment assigned to the patient at baseline (as randomized). FAS is the primary analysis set for efficacy endpoints.

## 3.2. The Per Protocol Set (PPS)

The per protocol set (PPS) includes all patients in the FAS who had a baseline and at least 1 post-baseline assessment of BCVA, and did not have any relevant important protocol violations that affect the primary efficacy variable. The final determination on the exclusion of patients from the PPS will be made on the masked data prior to the first database lock and described in a separate document. The PPS will be used for supplementary analysis of change from baseline in BCVA (non-inferiority only) at week 48 (primary endpoint) and week 60 (key secondary endpoint).

Treatment assignment is based on the treatment received (as treated). In general, the randomized treatment group will be considered as the actual treatment group, unless the patient has not been treated at all after randomization. Isolated incorrect treatments will not constitute a change in the "as treated" assignment but will be considered as intercurrent events (refer to Section 5.6.1).

## 3.3. The Safety Analysis Set (SAF)

The safety analysis set (SAF) includes all randomized patients who received any study treatment; it is based on the treatment received (as treated). Treatment compliance/administration and all clinical safety variables will be analyzed using the SAF. The safety analysis will be performed on the observed safety data.

## 3.4. Pharmacokinetic Analysis Sets

Two PK analysis sets will be defined. The PK analysis set (PKAS) includes all patients who received any study treatment and who had at least 1 non-missing PK result following the first dose of study drug. Patients will be analyzed based on actual treatment received.

The dense PK analysis set (DPKS) includes all patients who did not meet any of the additional exclusion criteria for Dense PK substudy who consented to Dense PK sampling (enrolled in PK sub study), received any study treatment, and with at least 1 non-missing dense PK result post first dose. Patients will be analyzed based on actual treatment received.

## 3.5. Immunogenicity Analysis Sets

The ADA analysis set (AAS) includes all treated patients and had at least 1 non-missing result in the ADA assay following the first study dose. Samples positive in the ADA assay will be analyzed in the Neutralizing antibody (NAb) assay.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

The NAb analysis set (NAbAS) includes all treated patients that are included in the ADA analysis set and that tested negative at all ADA sampling times or tested positive at one or more post-dose ADA sampling times and had at least one non-missing post-dose NAb result (either imputed or analysis result). Samples that tested negative for ADA are not assayed in the NAb assay and the corresponding NAb result are imputed as negative and included as such in the NAb analysis set. Patients in the NAbAS with multiple post-dose ADA results which consist of both imputed NAb-negative result(s) for ADA negative samples and only missing NAb results for all ADA-positive result(s), are set to NAb negative. Patients in the NAbAS that have at least one post-dose positive NAb analysis result are set to NAb positive even if other NAb results are missing.

#### 4. ANALYSIS VARIABLES

## 4.1. Demographic and Baseline Characteristics

The following demographic variables and baseline assessments will be summarized:

- Age
- Age category (<55 years,  $\ge55$  years to <65 years,  $\ge65$  years to <75 years,  $\ge75$  years)

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

- Sex (Female, Male)
- Race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Other, Not Reported)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not Reported)
- Geographical region (Japan, Rest of World).
- Weight (kg)
- Height (cm)
- Body mass index (BMI) (kg/m²)
- BMI category ( $\leq 30 \text{ kg/m}^2$ ,  $> 30 \text{ to } \leq 35 \text{ kg/m}^2$ ,  $> 35 \text{ kg/m}^2$ )
- Smoking history (Yes, No)
- Hemoglobin A1c (HbA1c)
- HbA1c category ( $\leq 8\%$ , > 8%)
- Vital Signs (heart rate, blood pressure [BP] [systolic and diastolic], and temperature)
- Intraocular pressure (IOP) in the study eye
- Medical history: renal impairment (Normal, Mild, Moderate, Severe), hepatic impairment (Yes, No), hypertension (Yes, No), cerebrovascular disease (Yes, No), ischaemic heart disease (Yes, No). Detailed definitions are presented in Appendix 10.4.
- Duration of diabetes (years): defined as time from diagnosis (based on medical history data (MedDRA High Level Term (HLT) "diabetes mellitus") to randomization
- Diabetes type (Type 1, Type 2)
- Diabetic Retinopathy Severity Scale (DRSS) in the study eye
- BCVA (measured by Early Treatment Diabetic Retinopathy Study [ETDRS] letters) in the study eye
- BCVA category (≤73 letters, >73 letters)
- CRT in the study eye
- Categorized CRT ( $<400 \mu m$ ,  $\ge 400 \mu m$ )


- National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) total score
- Prior DME treatment in the study eye (Yes, No)
- Presence of Clinically Significant Macular Edema (CSME)

## 4.2. Medical History

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA®).

#### 4.3. Pre-Treatment / Concomitant Medication

Medications taken during the study will be recorded and will be coded using the World Health Organization Drug Dictionary (WHODD).

Medications will be summarized as follows:

- **Prior medication** is defined as medication that was started before a patient received first study treatment regardless of when it was stopped.
- Concomitant medication is defined as medication that was ongoing at, or began after, the start of study treatment

## 4.4. Exposure, Compliance, Additional Treatment to Study Treatment

#### **Exposure**

For each patient, the following variables will be used to examine exposure to study treatment for the study eye:

- Total number of active injections through weeks 48, 60, and 96
- Total number of sham injections through weeks 48, 60, and 96
- Duration of treatment calculated (Weeks) as: [(last study treatment [active or sham] date) (first study treatment [active or sham] date) + 28]/7 (28 days are added because of the minimum 4-week dosing interval in the study)
- Proportion of patients in HDq16 group maintaining q16 dosing interval or longer through weeks 48, 60, and 96
- Proportion of patients in HDq12 and HDq16 groups maintaining q12 dosing interval or longer through weeks 48, 60, and 96
- Proportion of patients in HDq12 and HDq16 groups with q12 or q16 or longer dosing interval as the last intended dosing interval at week 48, week 60, and week 96
- Proportion of patients in HDq12 and HDq16 groups shortening dosing interval to q8 at week 16 or week 20
- Proportion of HDq12 and HDq16 patients with a shortened dosing interval anytime through weeks 48, 60 and 96

The following variables will be used to evaluate the fellow eye treatment

- Total number of aflibercept injections
- Duration of fellow eye treatment calculated (Weeks) as: [(last fellow eye treatment date) (first fellow eye treatment date) + 28]/7 (28 days are added because of the minimum 4-week dosing interval in the fellow eye in the study)

#### **Compliance**

Compliance with protocol-defined study treatments (active and sham) from baseline through the following time points will be assessed per patient: 48 weeks, 60 weeks and 96 weeks will be calculated as follows:

Treatment Compliance = (Number of received injections [sham or active] through a given time period)/(Number of planned injections [sham or active] during period of participation in the study through the given time period)  $\times 100\%$ 

For the calculation of compliance all injections (regardless if they were sham or active) will be used.

## 4.5. Efficacy Variable

#### 4.5.1. Primary Efficacy Variable (s)

The primary efficacy variable is the change from baseline in BCVA (as measured by ETDRS letter score) at week 48.

## 4.5.2. Key Secondary Efficacy Variable(s)

The key secondary efficacy endpoints are:

- Proportion of patients with a  $\geq 2$  step improvement in DRSS at week 48
- Change from baseline in BCVA at week 60 (for EMA/PMDA [European Medicines Agency/Pharmaceuticals and Medical Devices Agency] Analysis Plan only, see Section 5.6)

#### 4.5.3. Additional Secondary Efficacy Variable(s)

The additional secondary efficacy endpoints are:

Proportion of patients gaining  $\geq 15$  letters in BCVA from baseline at week 48

- Proportion of patients with BCVA  $\geq$  69 letters at week 48
- Proportion of patients without fluid at foveal center at week 48
- Change from baseline in CRT at week 48
- Proportion of patients without leakage on fluorescein angiography (FA) at week 48
- Change from baseline in NEI-VFQ-25 total score at week 48 (scoring details can be found in Appendix 10.3)

#### 4.5.4. Exploratory Efficacy Variable(s)

The exploratory efficacy endpoints will include the following:

- Change from baseline in BCVA at week 96
- Proportion of patients gaining  $\geq$  15 letters in BCVA from baseline at week 60 and 96

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

- Proportion of patients with BCVA  $\geq$  69 letters at week 60 and 96
- Change from baseline in CRT at week 60 and 96
- Proportion of patients without leakage on FA at week 60 and 96
- Change from baseline in NEI-VFQ-25 total score at week 60 and 96
- Proportion of patients without retinal fluid (total fluid, intraretinal fluid [IRF], subretinal fluid [SRF]) at the foveal center and in center subfield at week 48, week 60, and week 96
- Time to fluid-free retina over 48 weeks, 60 weeks, and 96 weeks (total fluid, IRF, SRF at foveal center and in the center subfield)
- Proportion of patients with sustained fluid-free retina (defined as the absence of fluid for at least 2 consecutive visits and for all subsequent study visits) over 48 weeks, 60 weeks, and 96 weeks (total fluid, IRF, SRF at foveal center and in the center subfield)
  - Sustained fluid-free retina is defined as the absence of fluid for at least 2 consecutive visits and for all subsequent study visits. The first 2 consecutive visits cannot have missing assessment between these two consecutive visits. After the 2 consecutive visits, the missing assessments at subsequent visits can be ignored or treated them as dry when determined sustained fluid free retina.
- Time to sustained fluid-free retina over 48 weeks, 60 weeks, and 96 weeks (total fluid, IRF, SRF at foveal center and in the center subfield)
- Proportion of patients without CSME at week 48, week 60, and week 96
- Proportion of patients with  $a \ge 3$  step improvement in DRSS at week 48, week 60, and week 96
- Change from baseline in BCVA averaged over the period from Week 36 to Week 48
- Change from baseline in BCVA average over the period from Week 48 to Week 60
- Proportions of patients gaining and losing  $\geq 5$  or  $\geq 10$  letters at week 48, week 60, and week 96
- Proportion of patients losing  $\geq$  15 letters at week 48, week 60, and week 96
- Proportion of patients randomized to HDq16 maintaining q16 dosing interval or longer through weeks 48, 60, and 96
- Proportion of patients randomized to HDq12 maintaining q12 dosing interval or longer through weeks 48, 60 and 96
- Proportion of patients with an assigned injection interval of  $\ge 16$  or  $\ge 20$  weeks based on assessment at the last injection visit (Week 96)

#### 4.6. Safety Variables

#### 4.6.1. Adverse Events and Serious Adverse Events

An adverse event (AE) is any untoward medical occurrence in a patient administered a study drug which may or may not have a causal relationship with the study drug.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

All AEs are to be coded according to MedDRA.

A Serious Adverse Event (SAE) is an AE that is classified as serious according to the criteria.

Other variables for AE description and analysis will include AE Verbatim Term, AE start date and end date/ongoing and corresponding study day, AE duration, relationship of AE to study drug, relationship of AE to 2 mg aflibercept in the fellow eye, relationship of AE to injection procedure, relationship of AE to study conduct, seriousness, severity, action due to AE, treatment of AE and outcome.

#### 4.6.2. Laboratory Safety Variables

The clinical laboratory data consists of serum chemistry, hematology, urinalysis and HbA1c.

Clinical laboratory values will be converted to standard international (SI) units and grouped by function in summary tables. Functions are defined as follows:

- Blood chemistry panel: Sodium, Potassium, Chloride, Carbon dioxide, Calcium, Glucose, Albumin, Total Protein (serum), Creatine, Blood urea nitrogen (BUN), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alkaline phosphatase, Lactate dehydrogenase (LDH), Total bilirubin, Total cholesterol (Low-density lipoprotein [LDL] + high-density lipoprotein [HDL]), Triglycerides, Uric acid, Creatine phosphokinase (CPK)
- Hematology panel: Hemoglobin, Hematocrit, Red blood cells (RBCs), White blood cells (WBCs), Red Cell Indices, Platelet count and Differential count (Neutrophils, Lymphocytes, Monocytes, Basophils, Eosinophils)
- Urinalysis: Color, Clarity, pH, Specific gravity, Ketones, Protein, Urine protein:creatinine ratio (UPCR), Glucose, Blood, Bilirubin, Leukocyte esterase, Nitrite, WBC, RBC, Hyaline and other casts, Bacteria, Epithelial cells, Crystals, Yeast
- HbA1c

#### 4.6.3. Vital Signs

Variables of analysis for vital signs include temperature, BP (systolic and diastolic) and heart rate.

#### 4.6.4. 12-Lead Electrocardiography (ECG)

Variables of 12-Lead Electrocardiogram (ECG) include PR interval, QRS interval, RR interval, QT interval, QTc with Fridericia corrections, and heart rate.

#### 4.6.5. Other Ocular Safety Variables

Other ocular safety variables include intraocular pressure pre-dose in the study eye and fellow eye and post-dose in the study eye.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

#### 4.6.6. Surgeries

All the surgeries after informed consent are collected on the case report form (CRF) and are coded by MedDRA. Treatment emergent surgery is defined as surgery performed during the ontreatment period (see Section 5.7.1).

#### 4.7. Pharmacokinetic Variables

The PK variables are the concentrations of free, bound, adjusted bound, and total aflibercept in plasma at each time point. Plasma samples for drug concentration will be collected at the clinic visits specified in the protocol schedule of events.

## 4.8. Immunogenicity Variables (ADA)

The immunogenicity variables include ADA status, NAb status and titer at nominal sampling time/visit. Serum samples for ADA will be collected at the clinic visits specified in Appendix 10.2.

#### 5. STATISTICAL METHODS

For continuous variables, descriptive statistics will include the following: the number of patients reflected in the calculation (n), mean, median, standard deviation, minimum, and maximum.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

For categorical or ordinal data, frequencies and percentages will be displayed for each category.

## **5.1.** Demographics and Baseline Characteristics

Demographic data and baseline characteristics variables will be summarized, by treatment group and overall, using descriptive statistics for FAS, SAF, and PPS. Disease characteristics of the study eye will be presented in a separate table.

## 5.2. Medical History

Medical history will be descriptively summarized, by treatment group and overall, for SAF. Summaries will show number and percentage of patients by primary system organ class (SOC) and preferred term (PT). The tables will be sorted by decreasing frequency of primary SOC. Within each primary SOC, PTs will be sorted by decreasing frequency in the total group. It will be summarized separately by ocular medical history in the study eye, ocular medical history in the fellow eye, and non-ocular medical history.

#### 5.3. Prior/concomitant Medications

All prior/concomitant medications, dictionary coded by WHODD, will be descriptively summarized by treatment group for SAF. Summaries will present number and percentage of patients for the medication groups described in Section 4.3 for all medications, by decreasing frequency of Anatomical Therapeutic Chemical (ATC) level 1 followed by ATC level 2 in the total group. In case of equal frequency across anatomic or therapeutic categories, alphabetical order will be used. Patients will be counted once in each ATC category (anatomic or therapeutic) linked to the medication.

Concomitant medications will be summarized by the following periods:

- Day 1 up to week 48
- Day 1 up to week 60
- Day 1 up to End of study (week 96)

When medication start/end date is missing, the rules for determining whether a medication is prior, concomitant, or post-treatment, are specified in Section 6.5.

## **5.4.** Patient Disposition

The disposition of patients in the study will be summarized by treatment group and overall. Percentages will be calculated using the number of randomized patients as the denominator. The following summaries will be provided:

- The total number of screened patients who have signed the ICF, the number of screen failure and the reasons for screen failure.
- The total number of randomized patients who received a randomization number


- The total number of patients in each analysis set
- The total number of patients who prematurely discontinued the study, and the reasons for discontinuation, and who completed the Week 48, Week 60, and Week 96 visits

## **5.5.** Extent of Study Treatment Exposure and Compliance

The variables for dose exposure and compliance described in Section 4.4 will be summarized for the SAF, FAS, and PPS populations, using descriptive statistics by the following time periods:

- Day 1 to week 48 (excluding treatment at week 48)
- Day 1 to week 60 (excluding treatment at week 60)
- Day 1 to End of study (week 96)

## 5.6. Analyses of Efficacy Variables

Due to differing requirements for the submission to regulatory authorities, 2 different analysis strategies will be applied, which will be detailed in this SAP document: a global statistical analysis plan (G-SAP), and a plan that specifically addresses requirements from EMA and PMDA (EP-SAP). The G-SAP will constitute the primary analysis for the study. The EP-SAP will be used for submission to the EMA/PMDA regulatory authorities.

All efficacy analyses will be conducted using the FAS population. In addition, the change from baseline in BCVA at week 48 and week 60 will be analyzed using the PPS population as supplementary analyses.

#### **5.6.1.** Analysis of Primary Efficacy Variable

The primary analysis is based on the estimand concept. The estimand of primary interest will be based mainly on a hypothetical strategy (ICH E9 [R1], 2017). It describes the change from baseline for all patients who started treatment, assuming all patients have stayed on treatment until week 48.

The estimand is specified through the following definitions of population, variable, treatment condition, intercurrent events, and population-level summary:

- Population: Defined by the inclusion/exclusion criteria. All efficacy analyses will be conducted using the FAS.
- Variable: Change from baseline to week 48 in BCVA
- Treatment condition: Intention to treat with HD aflibercept administered every 12 weeks (HDq12) after 3 initial monthly injections or every 16 weeks (HDq16) after 3 initial monthly injections each versus aflibercept 2 mg administered every 8 weeks (2q8) after 5 initial monthly injections; dose regimen modifications as detailed in Section 2.1 do not affect patient's assigned ITT regimen.
- Intercurrent events: Premature discontinuation from treatment; missed injections; use of prohibited medication; wrong study intervention administered, as displayed in Table 1.

Date: 19 AUGUST 2022 in least-square (LS) mean change from baseline to

Protocol: VGFTe-HD-DME-1934

• Population-level summary: Difference in least-square (LS) mean change from baseline to week 48 in BCVA between HDq12 and 2q8 (and HDq16 and 2q8) resulting from a mixed-model for repeated measurements (MMRM).

**Table 1: Strategies for occurrence of intercurrent events (ICE)** 

| Potential post-<br>randomization event | Intercurrent<br>event<br>(yes/no) | Estimand strategy | Analysis strategy |
|---|---|---|---|
| Premature<br>discontinuation of study<br>intervention before<br>Week 48 | | | |
| - Discontinuation of study at the same time | Yes | Hypothetical | Non-observed data beyond discontinuation will be covered implicitly in the MMRM |
| <ul> <li>Continuation of<br/>study beyond<br/>discontinuation of<br/>study intervention^</li> </ul> | Yes | Hypothetical | Observed data beyond last active injection prior to discontinuation + current treatment interval + 5 days will be excluded from analysis. Missing and excluded data will be covered by the MMRM. |
| Missed injection for any reason before Week 48 | | | |
| - Planned to be sham | Yes, but no impact | N/A | All observed data will be included in the analysis |
| - Planned to be active,<br>make-up given at<br>next visit | Yes | Treatment policy | All observed data will be included in the analysis |
| - Planned to be active, make-up or scheduled active injection not given at next visit | Yes | Hypothetical | Observed data beyond last active injection prior to the missed dose + current treatment interval + 5 days will be excluded from analysis. Missing and excluded data will be covered by the MMRM. |
| Shortening of dosing interval according to DRM criteria before Week 48 | No, DRM is considered part of the treatment regimen | N/A | ř |

| Use of a prohibited medication after the first dose of study medication ( | Yes | Hypothetical | Observed data beyond first administration of prohibited medicine will be excluded from analysis. Missing and excluded data will be covered by the MMRM. |
|---|---|---|---|
| Wrong study | | | |
| intervention before | | | |
| Week 48 | | | |
| <ul> <li>Active injection given instead of sham</li> </ul> | Yes | Treatment policy | All observed data will be included in the analysis |
| - Sham injection instead of active | Yes | Hypothetical | Observed data beyond last active injection prior to the wrong dose + current treatment interval + 5 days will be excluded from analysis. Missing and excluded data will be covered by the MMRM. |
| - Wrong dose level<br>given (eg, 2mg<br>given instead of<br>8mg) | Yes | Treatment policy | All observed data will be included in the analysis |

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

The following 2 hypotheses will be tested in the primary analysis:

• HDq12 is non-inferior to 2q8 regarding the mean change in BCVA from baseline to week 48 using a non-inferiority margin of 4 letters:

 $H_{10}$ :  $\mu_1 \le \mu_0 - 4$  vs.  $H_{11}$ :  $\mu_1 > \mu_0 - 4$ , where  $\mu_0$ ,  $\mu_1$ , are the mean change from baseline in BCVA at week 48 for 2q8 and HDq12, respectively.

• HDq16 is non-inferior to 2q8 regarding the mean change in BCVA from baseline to week 48 using a non-inferiority margin of 4 letters:

 $H_{30}\colon\ \mu_2\leq\mu_0-4\ vs.\ H_{31}\colon\ \mu_2>\mu_0-4,$ 

where  $\mu_0$ ,  $\mu_2$  are the mean change from baseline in BCVA at week 48 for 2q8, and HDq16, respectively.

#### 5.6.1.1. Primary Analysis for Primary Efficacy Variable

For the analysis of the primary efficacy variable, a mixed model for repeated measurements (MMRM) will be used with baseline BCVA measurement as a covariate and treatment group (HDq16 vs. 2q8 and HDq12 vs. 2q8) and baseline CRT category (<400 μm, ≥400 μm), prior

<sup>^</sup> This ICE will be handled in the same way as "Missed injection: Planned to be active, make-up or scheduled active injection not given at next visit, since the info of discontinuation from study intervention was not collected in the database.

DME treatment (yes, no), geographical region (Rest of world, Japan), and visit as fixed effects as well as terms for the interaction between baseline BCVA and visit and for the interaction between treatment and visit. A Kenward-Roger approximation will be used for the denominator degrees of freedom. Further, an unstructured covariance structure will be used. If the model does not converge, an appropriate covariance structure will be used instead. Only data up to Week 48 will be used in this analysis.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

$$Y_{ijk} = \beta_0 + \beta_{baseBCVA} x_i + \beta_{treat}^{(k)} + \beta_{base\_CRT}^{(n)} + \beta_{pDME}^{(l)} + \beta_{reg}^{(m)} + \beta_{visit}^{(j)} + \beta_{treat*visit}^{(k,j)} + \beta_{base*visit}^{(j)} x_i + \epsilon_{ijk},$$

where:

 $Y_{ijk}$  is the change from baseline BCVA for  $i^{th}$ patient at  $j^{th}$ visit for  $k^{th}$  treatment group,  $\beta_0$  is an intercept term,

 $\beta_{baseBCVA}$  is the regression coefficient of the covariate,

 $x_i$  for the baseline BCVA of  $i^{th}$  patient,

 $\beta_{treat}^{(k)}$  is the fixed effect of treatment group k

 $\beta_{base\_CRT}^{(n)}$  is the fixed effect of categorized baseline CRT n,

 $\beta_{pDME}^{(l)}$  is the fixed effect of prior DME treatment l,

 $\beta_{reg}^{(m)}$  is the fixed effect of region m,

 $\beta_{visit}^{(j)}$  is the fixed effect of visit j,

 $\beta_{base*visit}^{(j)}$  the interaction between baseline BCVA and visit j,

 $\beta_{treat*visit}^{(k,j)}$  the interaction between treatment k and visit j,

 $\epsilon_{ijk}$  is the residual error with  $\epsilon_{ijk} \sim N(0, \sigma^2)$  and  $corr(\epsilon_{ijk}, \epsilon_{ij'k}) = \rho^{(k)} \{i, j'\}$ , or 0 otherwise.

In terms of the estimators the population-level summary of the estimands (ie, the treatment effect at week 48) can then be expressed as

$$D_{HDQ12} = \left[\beta_{treat}^{(HDQ12)} + \beta_{treat*visit}^{(HDQ12,w48)}\right] - \left[\beta_{treat}^{(2Q8)} + \beta_{treat*visit}^{(2Q8,w48)}\right]$$

and

$$D_{HDQ16} = \left[\beta_{treat}^{(HDQ16)} + \beta_{treat*visit}^{(HDQ16,w48)}\right] - \left[\beta_{treat}^{(2Q8)} + \beta_{treat*visit}^{(2Q8,w48)}\right].$$

Summary tables will include number of patients, LS mean change, (unadjusted) mean change and standard deviation (SD) and baseline means of each treatment group. For non-inferiority testing, the population level estimates comparing HDq16 vs. 2q8 ( $D_{HDQ16}$ ) and HDq12 vs. 2q8 ( $D_{HDQ12}$ ), expressed as LS mean change, the test statistics, the degrees of freedom, and

corresponding p-values will be presented. Two-sided 95% confidence intervals will also be provided.

In line with the definition of estimands (see above), the primary analysis will be performed on the FAS and patients will be analyzed within their original randomized group (regardless of any changes to dose interval). The MMRM assumes missing at random (MAR) for patients who discontinue the study prematurely, ie, missingness only depends on observed data.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

The following superiority testings will be performed as described in Section 5.6.4 for G-SAP strategy and EP-SAP strategy.

• HDq12 is superior to 2q8 regarding the mean change in BCVA from baseline to week 48:

 $H_{70}$ :  $\mu_1 \le \mu_0$  vs.  $H_{71}$ :  $\mu_1 > \mu_0$ , where  $\mu_0$ ,  $\mu_1$ , are the mean change from baseline in BCVA at week 48 for 2q8 and HDq12, respectively.

• HDq16 is superior to 2q8 regarding the mean change in BCVA from baseline to week 48:

 $H_{90}$ :  $\mu_2 \le \mu_0 \text{ vs. } H_{91}$ :  $\mu_2 > \mu_0$ ,

where  $\mu_0$ ,  $\mu_2$  are the mean change from baseline in BCVA at week 48 for 2q8, and HDq16, respectively.

An example of Statistical Analysis System (SAS) code for MMRM is presented in Appendix 10.8

#### 5.6.1.2. Sensitivity Analyses for Primary Efficacy Variable

Last observation carried forward (LOCF) will be conducted for patients who had at least one post-baseline value but discontinued prematurely or had an ICE as defined in Table 1 before week 48 and ANCOVA will be applied for the change from baseline in BCVA at week 48. Another approach assuming MAR will be implemented by using multiple imputation (MI). In addition, the tipping point analysis will be performed as a sensitivity analysis if the MI analysis results under MAR assumption show non-inferiority of the high dose groups compared to the low dose group.

#### 5.6.1.2.1. ANCOVA using LOCF

For this sensitivity analysis of the primary efficacy variable, an analysis of covariance (ANCOVA) will be used with baseline BCVA measurement as a covariate and treatment group (HDq16 vs. 2q8 and HDq12 vs. 2q8) and the stratification variables (baseline CRT category [<400  $\mu$ m,  $\geq$ 400  $\mu$ m], prior DME treatment [yes, no], geographical region [Rest of world, Japan]) as fixed factors. A separate variance term will be estimated for the three treatment groups.

The observation at week 48 of patient *i* receiving treatment *t* can be written as follows:

$$Y_{itrb} = \mu_t + \gamma_r + \eta_c + \pi_n + x_i \beta + \epsilon_{itrb}$$

where

Y<sub>itrh</sub> is the change from baseline to week 48 for the *i*th patient,


 $\mu_t$  is the treatment effect,

 $\gamma_r$  is the geographic region effect (Rest of world, Japan),

 $\eta_c$  is the categorized baseline CRT (<400 µm,  $\geq$ 400 µm),

 $\pi_p$  is the prior DME treatment (yes, no)

 $x_i$  is the baseline BCVA of patient i,

 $\epsilon_{itrb}$  is the residual error with  $\epsilon_{itrb} \sim N(0, \sigma_t^2)$  for treatment arm t.

For this analysis missing week 48 BCVA data will be imputed by using LOCF. That means that the last non-missing post-baseline BCVA measurement prior to an ICE will be carried forward to week 48.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

Summary tables will include number of patients, LS mean change, (unadjusted) mean change and SD and baseline means of each treatment group. For non-inferiority testing the one-sided  $\alpha$  of 0.025 for the population level estimates comparing HDq16 vs. 2q8 and HDq12 vs. 2q8, the estimates expressed as LS mean change including the one-sided confidence intervals (CIs) for  $\alpha$  of 0.025, the test statistics, the degrees of freedom and corresponding p-values will be presented.

This sensitivity analysis will be analyzed for the FAS.

An example of SAS code for ANCOVA is presented in Appendix 10.8.

#### 5.6.1.2.2. ANCOVA with Multiple Imputation

The primary efficacy variable at week 48 will be analyzed using MI with ANCOVA model based on the FAS. Data after occurrence of an ICE as defined in Table 1 will be excluded. MI methods involve three steps.

#### I. Imputation

Missing data up to week 48 will be imputed 50 times to generate 50 complete data sets by using the SAS procedure MI following the 2 steps below:

<u>Step 1</u>: The monotone missing pattern is induced by Markov Chain Monte Carlo (MCMC) method in MI procedure using seed number 01934.

Step 2: The missing data at subsequent visits will be imputed using the regression method for the monotone pattern with seed number 01934 and adjustment for covariates including treatment groups, baseline CRT category ( $<400 \mu m$ ,  $\ge 400 \mu m$ ), prior DME treatment (yes, no), geographical region (Rest of world, Japan), baseline BCVA and all BCVA values at preceding visits.

If the imputed data is outside the range of 0 to 100 in either step of imputation, truncation will be applied to the imputed data.

#### II. Analysis

The week 48 data of each of the 50 complete datasets will be analyzed using an ANCOVA model as specified in Section 5.6.2.2.1.

#### III. Pooling

The SAS MIANALYZE procedure will be used to generate valid statistical inferences by combining results from the 50 analyses using Rubin's formula (Rubin, 1987).

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

An example of SAS code for MI is presented in Appendix 10.8.

### 5.6.1.2.2.1. Tipping Point Analysis

In order to check the assumption that the missing data are not MAR, a tipping point analysis will be conducted based on the multiple imputation analysis in Section 5.6.1.2.2. The objective of the tipping point analyses is to identify assumptions about the missing data under which the conclusions from the main analysis change, ie, under which non-inferiority cannot be shown anymore. These tipping point analyses will only be performed if the multiple imputation analysis results show non-inferiority of the high dose groups compared to the low dose group. In case the non-inferiority is shown, additional tipping point analyses will be repeated after reducing the imputed BCVA values in the high dose arms by ascending natural number of letters (1, 2, 3... etc.), with the goal to find for each high dose treatment group the "tipping point" that will significantly reverse the analysis result. The smallest delta, for which non-inferiority cannot be shown anymore, will be the "tipping point".

For each value of delta, summary tables will include number of patients, LS mean change, (unadjusted) mean change and SD and baseline means of each treatment group as well as the estimates expressed as LS mean change including the two-sided CIs, the test statistics, the degrees of freedom and corresponding p-values.

An example of SAS code for tipping point analysis is presented in Appendix 10.8.

#### **5.6.1.3.** Supplementary Analyses for Primary Efficacy Variable

The primary analysis described in Section 5.6.1.1 will be repeated using the PPS.

#### **5.6.1.4.** Subgroup Analyses for Primary Efficacy Variable

Analyses will be performed in the following subgroups:

- Sex: male, female
- Age at enrollment: <55 years, ≥55 years to <65 years, ≥65 years to < 75 years, ≥75 years
- Race (only subgroups with sufficient sample size): White, Black or African American, Asian
- Ethnicity: Not Hispanic or Latino, Hispanic or Latino
- Baseline BCVA (≤73 letters, >73 letters)
- Geographic region: Japan, Rest of the world
- Baseline CRT category (<400 μm, ≥400 μm)
- Prior DME treatment (yes, no)

Subgroup analyses will be performed using the same model as in Section 5.6.1.1, except for those subgroups that are also stratification factors (geographic region, baseline CRT category,

and prior DME treatment), where these terms will be individually removed from the model (leaving the other 2 factors in).

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

#### 5.6.2. Analysis of Key Secondary Efficacy Variables

## 5.6.2.1. Change from Baseline in BCVA Measured by the ETDRS Letter Score at Week 60

The following 2 non-inferiority hypotheses will be tested for this key secondary endpoint under the EP-SAP only:

- HDq12 is non-inferior to 2q8 regarding the mean change in BCVA from baseline to week 60 using a non-inferiority margin of 4 letters:
  - $H_{20}$ :  $\mu_1 \le \mu_0 4$  vs.  $H_{21}$ :  $\mu_1 > \mu_0 4$ ,
  - where  $\mu_0$ ,  $\mu_1$ , are the mean change from baseline in BCVA at week 60 for 2q8 and HDq12, respectively.
- HDq16 is non-inferior to 2q8 regarding the mean change in BCVA from baseline to week 60 using a non-inferiority margin of 4 letters:
  - $H_{40}$ :  $\mu_2 \le \mu_0 4 \text{ vs. } H_{41}$ :  $\mu_2 > \mu_0 4$ ,
  - where  $\mu_0$ ,  $\mu_2$  are the mean change from baseline in BCVA at week 60 for 2q8, and HDq16, respectively.

The analysis of key secondary endpoints will be required for the submission to the EMA/PMDA regulatory authorities. The change from baseline in BCVA at week 60 will be analyzed with the same methods and main and sensitivity summaries as for the primary endpoint described in Section 5.6.1. Only data up to Week 60 will be used in this analysis.

The following superiority testings will also be performed as described in Section 5.6.4 (under the EP-SAP only) for this endpoint.

- HDq12 is superior to 2q8 regarding the mean change in BCVA from baseline to week 60:  $H_{80}$ :  $\mu_1 \le \mu_0$  vs.  $H_{81}$ :  $\mu_1 > \mu_0$ , where  $\mu_0$ ,  $\mu_1$ , are the mean change from baseline in BCVA at week 48 for 2q8 and HDq12, respectively.
- HDq16 is superior to 2q8 regarding the mean change in BCVA from baseline to week 60:  $H_{100}$ :  $\mu_2 \le \mu_0$  vs.  $H_{101}$ :  $\mu_2 > \mu_0$ , where  $\mu_0$ ,  $\mu_2$  are the mean change from baseline in BCVA at week 48 for 2q8, and HDq16, respectively.

Subgroup analyses will be performed on those subgroups listed in Section 5.6.1.4 using the same model described above, except for those subgroups that are also stratification factors (geographic region, baseline CRT category, and prior DME treatment), where these terms will be individually removed from the model (leaving the other 2 factors in).

#### 5.6.2.2. Proportion of patients with a $\geq$ 2 step improvement in DRSS at week 48

The following 2 non-inferiority hypotheses will be tested for this key secondary variable on the FAS:

• HDq12 is non-inferior to 2q8 regarding the proportion of patients with a ≥2 step improvement in DRSS at week 48:

```
H<sub>50</sub>: p_{HDq12} \le p_{2Q8} - 0.15 vs. H<sub>51</sub>: p_{HDq12} > p_{2Q8} - 0.15, where p_{2Q8}, p_{HDq12}, are the proportion of patients with a \ge 2 step improvement in DRSS at week 48 for 2q8, and HDq12, respectively.
```

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

• HDq16 is non-inferior to 2q8 regarding the proportion of patients with a ≥2 step improvement in DRSS at week 48:

```
H<sub>60</sub>: p_{HDq16} \le p_{2Q8} - 0.15 vs. H<sub>61</sub>: p_{HDq16} > p_{2Q8} - 0.15, where p_{2Q8}, p_{HDq16}, are the proportion of patients with a \ge 2 step improvement in DRSS at week 48 for 2q8, and HDq16, respectively.
```

The non-inferiority margin is set at 15%. This endpoint will be analyzed by a Cochran-Mantel-Haenszel (CMH) test stratified by baseline CRT category ( $<400~\mu m, \ge 400~\mu m$ ), prior DME treatment (yes, no), geographical region (Rest of world, Japan). Missing or non-gradable post-baseline values will be imputed using LOCF procedure. Patients will be considered as non-responders if all post-baseline measurements are missing or non-gradable. Strategies for occurrence of intercurrent events will be similar to Table 1, except the excluded data will be implemented by LOCF procedure.

Additionally, a two-sided 95% Mantel-Haenszel confidence interval (Koch et al, 1990) for the difference of proportion adjusted for stratification factors (baseline CRT category [<400 μm, ≥400 μm], prior DME treatment [yes, no], geographical region [Rest of world, Japan]) will be calculated using normal approximation.

Subgroup analyses will be performed on those subgroups listed in Section 5.6.1.4 using the same model described above, except for those subgroups that are also stratification factors (geographic region, baseline CRT category, and prior DME treatment), where these terms will be individually removed from the model (leaving the other 2 factors in).

#### **5.6.2.2.1.** Sensitivity Analyses

The following sensitivity analysis will be performed for the proportion of patients with a  $\geq$ 2 step improvement in DRSS at week 48 for the FAS:

The above analysis will be repeated but for observed cases (OC) only, ie, observed data prior to the occurrence of an ICE.

#### 5.6.3. Analysis of Additional Secondary and Exploratory Efficacy Variables

All additional secondary and exploratory efficacy variables (see Section 4.5.3 and Section 4.5.4) will be analyzed descriptively at each scheduled visit from baseline to week 48, week 60, and week 96, as applicable. These descriptive analyses will include statistical tests (with nominal p-values) for the efficacy variables and two-sided 95% confidence intervals.

For these statistical tests, continuous variables will be analyzed by the same repeated measurement models as for the primary endpoint.

Binary endpoints will be analyzed by CMH methods adjusted by the stratification factors based on LOCF (ie, missing/non-gradable data will be imputed by the last valid data prior to ICE). The endpoint of proportion of patients with  $a \ge 3$  step improvement in DRSS will analyzed by the

same method as the proportion of patients with  $a \ge 2$  step improvement in DRSS as specified in Section 5.6.2.2. For the other binary endpoints, only valid data (excluding missing/non-gradable) will be included in the denominator when calculated the proportion. Sensitivity analysis will be performed by OC method (ie, observed data prior to an ICE).

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

Time-to-event variables will be analyzed using the Kaplan-Meier method. Time to event will be calculated as duration from date of randomization to the event for the first time whereas intercurrent events are handled according to Table 1. Patients without the event will be censored at their last assessment date. The analysis will be using the study visits (ie, multiples of 4 weeks) and not the calendar time as unit. Each of the HD groups will be compared with the 2q8 group using a stratified log-rank test. Hazard ratios will be calculated using a stratified Cox proportional hazards model, including treatment group as factor and baseline CRT category (<400  $\mu$ m,  $\geq$ 400  $\mu$ m), prior DME treatment (yes, no), geographical region (Rest of world, Japan) as strata.

No multiplicity adjustments will be made for these efficacy analyses.

#### 5.6.4. Adjustment for Multiple Comparisons

For the G-SAP strategy, statistical hypotheses of the primary endpoint (BCVA at week 48) and the key secondary endpoint (≥2 step improvement in DRSS at week 48) will be assessed together, after all patients completed week 48 (or discontinued prematurely) using the below described methods.

For the EP-SAP strategy, statistical hypotheses of the primary endpoint (BCVA at week 48) and the key secondary endpoints (BCVA at week 60, ≥2 step improvement in DRSS at week 48) will be assessed together, after all patients completed week 60 (or prematurely discontinued) using the below described methods.

The overall family-wise type 1 error will be controlled at 0.025 (one-sided tests) for testing the primary and key secondary endpoints. Adjustment for multiple comparisons in the primary and key secondary endpoints will be made with a hierarchical testing procedure. This approach allows the confirmatory testing of a hypothesis at the full alpha level of 0.025 after successful rejection of the hypotheses which are ranked higher in the hierarchy. The hypotheses will be tested in the order as specified in Table 2 for G-SAP and EP-SAP, respectively.

Table 2: The Testing Order of Hierarchical Testing Procedure in G-SAP and EP-SAP

| G-SAP | EP-SAP |
|---|---|
| H <sub>10</sub> : Q12 BCVA Week 48 non-inferiority | H <sub>10</sub> : Q12 BCVA Week 48 non-inferiority |
| | H <sub>20</sub> : Q12 BCVA Week 60 non-inferiority |
| H <sub>30</sub> : Q16 BCVA Week 48 non-inferiority | H <sub>30</sub> : Q16 BCVA Week 48 non-inferiority |
| | H <sub>40</sub> : Q16 BCVA Week 60 non-inferiority |
| H <sub>50</sub> : Q12 DRSS Week 48 non-inferiority | H <sub>50</sub> : Q12 DRSS Week 48 non-inferiority |

| H <sub>60</sub> : Q16 DRSS Week 48 non-inferiority | H <sub>60</sub> : Q16 DRSS Week 48 non-inferiority |
|---|---|
| H <sub>70</sub> : Q12 BCVA Week 48 superiority | H <sub>70</sub> : Q12 BCVA Week 48 superiority |
| | H <sub>80</sub> : Q12 BCVA Week 60 superiority |
| H <sub>90</sub> : Q16 BCVA Week 48 superiority | H <sub>90</sub> : Q16 BCVA Week 48 superiority |
| | H <sub>100</sub> : Q16 BCVA Week 60 superiority |

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

## 5.7. Analysis of Safety Data

The safety variables as defined in Section 4.6 will be analyzed on the SAF for the periods from baseline/day 1 through week 48, week 60 and the end of study (week 96). The summary of safety results will be presented for each treatment group. Data will not be imputed for the safety analysis.

#### 5.7.1. Adverse Events

**Period of observation:** The observation period will be divided into three segments:

- The pretreatment period is defined as the time from signing the ICF to before the first dose of study drug
- The on-treatment period (to determine treatment-emergent adverse events [TEAEs]) is defined as the time from the first dose of study drug to the last dose of study drug (active or sham) plus 30 days. In the week 48 (week 60) analysis, for patients who are still participating in the study (ie, have not been withdrawn), all AEs up through the date of that visit will be considered on-treatment.
- The post-treatment period is defined as after the end of the on-treatment period

TEAEs are defined as events that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period.

TEAEs will further be summarized by the following categories:

- Ocular TEAEs in the study eye
- Ocular TEAEs in the fellow eye
- Non-ocular TEAEs

The following TEAE categories will also be summarized as described for TEAEs:

- Study drug related TEAEs
- Injection related TEAEs
- Study conduct related TEAEs
- 2mg aflibercept in the fellow eye related TEAEs
- TEAEs leading to discontinuation


Regeneron Pharmaceuticals, Inc.

Protocol: VGFTe-HD-DME-1934
Statistical Analysis Plan

Date: 19 AUGUST 2022

- TEAEs by maximum severity
- TE SAEs
- Study drug related TE SAEs
- Injection related TE SAEs
- TE SAEs by maximum severity

Counts will be provided according to treatment group for each PT within each SOC. Percentages will be calculated using the number of patients from the SAF in each treatment group.

Primary SOCs will be sorted according to alphabetical order. Within each primary SOC, PTs will be sorted by alphabetical order as well. For tables presenting severity of events, the worst severity will be chosen for patients with multiple instances of the same event.

Treatment emergent APTC events (adjudicated), hypertension, intraocular inflammation, and nasal mucosal events will be tabulated. Detailed definitions for the latter 3 of these types of AEs are presented in Appendix 10.4. Please refer to APTC charter for more information for adjudication of APTC events.

The following study periods will be used for TEAE summaries:

- Day 1 to week 48
- Day 1 to week 60
- Day 1 to week 96

#### 5.7.1.1. Subgroup Analyses

Subgroup analyses in TEAE reporting will be performed for the following subgroups:

- Sex: male, female
- Age at enrollment: <55 years, ≥55 years to <65 years, ≥65 years to <75 years, ≥75 years
- Race (only subgroups with sufficient sample size): White, Black or African American, Asian
- Ethnicity: Not Hispanic or Latino, Hispanic or Latino
- Geographic region: Japan, Rest of the world
- Medical history of renal impairment
- Medical history of hepatic impairment
- Medical history of hypertension
- Medical history of cerebrovascular disease
- Medical history of ischaemic heart disease

The medical history subgroups are defined in more detail in Appendix 10.4.

Regeneron Pharmaceuticals, Inc.

Protocol: VGFTe-HD-DME-1934
Statistical Analysis Plan

Date: 19 AUGUST 2022

Summaries (by SOC and PT) of patients with each of the following types of TEAE will be provided for the above subgroups:

- Ocular TEAEs in the study eye
- Non-ocular TEAEs
- Serious ocular TEAEs in the study eye
- Serious non-ocular TEAEs

#### 5.7.2. Clinical Laboratory Measurements

Baseline clinical laboratory analytes and change from Baseline in clinical laboratory analytes to each scheduled assessment time will be summarized with descriptive statistics.

Shift tables based on baseline normal/abnormal and other tabular and graphical methods may be used to present the results for laboratory tests of interest.

Listings will be provided with flags indicating the out of normal range values.

Treatment-emergent high abnormalities are laboratory values that were normal or low at Baseline but high after treatment with study drug. Treatment-emergent high abnormalities will be summarized using SAF for patients who were normal or low at Baseline.

Treatment-emergent low abnormalities are laboratory values that were normal or high at Baseline but low after treatment with study drug. Treatment-emergent low abnormalities will be summarized using SAF for patients who were normal or high at Baseline.

A treatment-emergent potentially clinically significant value (PCSV) is a laboratory value that was normal at Baseline but met PCSV criteria after treatment with study drug. Definitions of PCSVs are listed in Appendix 10.5. Treatment Emergent PCSVs will be summarized using SAF for patients who did not meet the PCSV criterion at baseline.

#### 5.7.3. Analysis of Vital Signs

The assessments of vital signs (heart rate, systolic/diastolic BP, and temperature) and their changes from Baseline will be summarized by visit. The Baseline for BP is defined as the average of all valid measurements taken prior to administration of study drug. The Baseline for other vital signs endpoints will be the latest available valid measurement taken prior to the administration of study drug, as specified in 6.1.

Treatment Emergent PCSV for systolic/diastolic blood pressure will be summarized based on the using SAF and in the SAF for patients who do did not meet the PCSV criterion at baseline. Definition of PCSVs for blood pressure are listed in Appendix 10.5.

#### 5.7.4. Analysis of 12-Lead ECG

The assessments of ECG parameters (P-R interval, QT interval, QTc interval, QRS interval, Ventricular rate and Heart rate) and their changes from Baseline will be summarized by visit.

ECG status (ie, normal, abnormal) will be reported. Shift tables may be provided to present the post-baseline status according to the baseline status (normal or missing / abnormal) by treatment group.

#### 5.7.5. Analysis of Other Ocular Safety Variables

Pre-dose IOP measurements and their changes from baseline will be summarized by visit using descriptive statistics for the study eye and the fellow eye, respectively. Post-dose IOP measurements and their changes from pre-dose will be summarized for study eye. The proportion of patients who meet the following criteria will be summarized descriptively:

•  $\geq$  10 mmHg increase in IOP measurement from baseline to pre-dose measurement in the study eye (by visit and at any time)

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

- ≥ 10 mmHg increase in IOP measurement from baseline to pre-dose measurement in the fellow eye (by visit and at any time)
- > 21 mmHg for any pre-dose measurement in the study eye (by visit and at any time)
- > 21 mmHg for any pre-dose measurement in the fellow eye (by visit and at any time)
- $\geq$  25 mmHg for any pre-dose measurement in the study eye (by visit and at any time)
- $\geq$  25 mmHg for any pre-dose measurement in the fellow eye (by visit and at any time)
- $\geq$  35 mmHg at any time (pre- or post-dose) in the study eye (by visit and at any time)
- $\geq$  35 mmHg at any time (pre- or post-dose) in the fellow eye (by visit and at any time)

#### 5.7.6. Surgeries

Treatment emergent surgeries will be summarized by the following categories:

- Ocular treatment emergent surgeries in the study eye
- Ocular treatment emergent surgeries in the fellow eye
- Non-ocular treatment emergent surgeries

## 5.8. Analysis of Pharmacokinetic Data

#### 5.8.1. Analysis of Drug Concentration Data

#### **Main Study:**

The concentrations of free, bound, adjusted bound, and total aflibercept over time will be summarized by descriptive statistics for each treatment group. Concentrations may be further grouped by factors such as age, renal function, HbA1c level, hepatic function, concomitant medications, body weight, ethnicity, etc. No formal statistical hypothesis testing will be performed.

#### **Dense PK Substudy:**

The PK parameters to be determined after the first dose for free, adjusted bound, and total aflibercept may include, but are not limited to:

- C<sub>max</sub>
- C<sub>max</sub>/Dose
- $\bullet$   $t_{max}$

Regeneron Pharmaceuticals, Inc. Statistical Analysis Plan

- t<sub>last</sub>
- C<sub>last</sub>
- AUC<sub>last</sub>
- AUCinf
- AUCinf/Dose
- t<sub>1/2</sub>
- C<sub>trough</sub>

After repeat dosing in the dense PK substudy, PK parameters to be determined may include, but are not limited to, C<sub>trough</sub>, time to reach steady-state, and accumulation ratio. PK parameters will be summarized by descriptive statistics by treatment group, and geographical region as appropriate. This descriptive statistical assessment may include the geometric means and ratios of the geometric means for selected PK parameters, as deemed appropriate. No formal statistical hypothesis testing will be performed.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

#### **5.8.2.** Pharmacokinetics/Pharmacodynamics Analyses

Dose- and/or exposure-response analyses for efficacy and safety endpoints may be performed, as appropriate.

### 5.9. Analysis of Immunogenicity Data

The immunogenicity variables described in Section 4.8 will be summarized using descriptive statistics. Immunogenicity will be characterized per drug molecule by ADA status, ADA category and maximum titer observed in patients in the ADA analysis sets.

The ADA status of each patient may be classified as one of the following:

- Positive
- Pre-existing If the baseline sample is positive and all post baseline ADA titers are reported as less than 4-fold the baseline titer value
- Negative If all samples are found to be negative in the ADA assay.

The ADA category of each positive patient is classified as:

Treatment-boosted - A positive result at baseline in the ADA assay with at least one post baseline titer result ≥4-fold the baseline titer value

Treatment-emergent - A negative result or missing result at baseline with at least one positive post baseline result in the ADA assay. Patients that are treatment-emergent will be further categorized as follows:

Persistent - A positive result in the ADA assay detected in at least 2 consecutive post baseline samples separated by at least a 16-week post baseline period [based on nominal sampling time], with no ADA-negative results in-between, regardless of any missing samples

Transient - Not persistent or indeterminate, regardless of any missing samples


Indeterminate - A positive result in the ADA assay at the last collection time point only, regardless of any missing samples

The maximum titer category of each patient is classified as:

Low (titer < 1,000)

Moderate  $(1,000 \le \text{titer} \le 10,000)$ 

High (titer >10,000)

The following will be summarized by treatment group and ADA titer level:

Number (n) and percent (%) of ADA-negative patients

Number (n) and percent (%) of pre-existing patients

Number (n) and percent (%) of treatment-emergent ADA positive patients

#### 6. DATA CONVENTIONS

The following analysis conventions will be used in the statistical analysis.

#### **6.1.** Definition of Baseline

Unless otherwise specified, the Baseline assessment for all measurements will be the latest available valid measurement taken prior to the administration of study drug.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

### 6.2. Visit Windows

The visits used for the analysis will be based on the nominal visits, ie, according to the case report form (CRF) assessment recorded by the investigator. No visit windows will be further defined.

#### 6.3. Unscheduled Assessments

Unscheduled assessments will not be included in the summaries unless specified.

If more than one value is available for a given visit, the visit value actually used for statistical summaries and analyses will be as follows:

- The last non-missing repeated measurement, if respective visit is before start of treatment
- The first non-missing repeated measurement, if respective visit is after start of treatment

If an early termination visit is performed within the protocol-defined window of the next scheduled visit after the last previous visit, the visit-dependent assessments will be re-slotted to the next scheduled visit.

## 6.4. Handling of Patients who Discontinue

Patients who discontinue this study will not be replaced. The details for the handling of missing data due to patients who discontinue the study and study medication are described in Section 6.5.

## 6.5. Data Handling Convention for Missing Data

For the primary and secondary efficacy variables, missing observations will be dealt with as described in the efficacy analysis (Section 5.6) based on the analysis being performed.

#### Pretreatment/concomitant medication

For the tabulation of prior and concomitant medication, partially missing start dates of the medication will be imputed by the earliest possible time point, partially missing stop dates will be imputed by the latest possible time point.

#### Adverse event

It is important to determine whether AEs started during the on-treatment period. AEs with partial start dates will be imputed based on the following rules:

1. If AE partial start date indicates it is before the first dose of study drug, then it will be imputed as the latest possible date

Regeneron Pharmaceuticals, Inc. Statistical Analysis Plan

Protocol: VGFTe-HD-DME-1934 Date: 19 AUGUST 2022

- 2. If AE partial start date has the same partial date as the first dose of study drug, then it will be imputed as the date of the first dose of study drug
- 3. If AE partial start date indicates it is after the first dose of study drug, then it will be imputed as the earliest possible date.
- 4. If imputed AE start date is later than AE end date, then impute the AE start date to AE end date.

### 7. INTERIM ANALYSIS

No formal interim analyses will be performed. However, the primary analysis for this study will be performed once all patients reach week 48, with a subsequent analysis performed when all patients reach week 60. The study will continue through week 96.

Protocol: VGFTe-HD-DME-1934

#### 8. **SOFTWARE**

All analyses will be done using SAS Version 9.4 (or higher) or R version 3.5.1 (or higher).

#### 9. REFERENCES

1. ICH. (1998, February 5). ICH Harmonized tripartite guideline: Statistical principles for clinical trials (E9). International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use.

Protocol: VGFTe-HD-DME-1934

- 2. Brown DM, Schmidt-Erfurth U, Do DV, HolzFG, Boyer DS, Midena E, et al. Intravitreal aflibercept for diabetic macular edema: 100-week results from the VISTA and VIVID studies. Ophthalmology 2015;122(10):2044-52.
- 3. Bretz F, Maurer W, Brannath W, Posch M. A graphical approach to sequentially rejective multiple test procedures. Statistics in Medicine. 2009;28:586–604
- 4. Bretz F, Posch M, Glimm E, Klinglmueller F, Maurer W, Rohmeyer K. Graphical approaches for multiple comparison procedures using weighted Bonferroni, Simes, or parametric tests. Biom J 2011;Nov 53(6):894-913.
- 5. Huque M, Mushti S, Alosh M. Recycling of Significance Levels in Testing Multiple Hypotheses of Confirmatory Clinical Trials. In Biopharmaceutical Applied Statistics Symposium. Singapore: Springer; 2018:91-118.
- 6. Rohmeyer K, Klinglmueller F. gMCP: Graph Based Multiple Test Procedures. R package version 0.8. 10. URL http://CRAN.R-project.org/package=gMCP 2015.
- 7. ICH E9 (R1) (2017) Statistical Principles for Clinical Trials: Addendum: Estimands and Sensitivity Analysis in Clinical Trials
- 8. Koch GG, Carr GJ, Amara IA, Stokes ME, Uryniak TJ, 'Categorical Data Analysis' in Statistical methodology in the pharmaceutical sciences / edited by DA Berry, Marcel Dekker, 1990
- 9. Rubin D E. Multiple Imputation for Nonresponse in Surveys. Wiley. 1987

## 10. APPENDIX

## 10.1. Summary of Statistical Analyses

## **Efficacy Analysis:**

| Endpoint | Analysis<br>Populations | Primary<br>Analysis | Statistical<br>Method | Supportive<br>Analysis | Subgroup<br>Analysis | Other<br>Analyses |
|---|---|---|---|---|---|---|
| Primary Endpoint | | | | | | |
| Change from<br>baseline in BCVA<br>at Week 48 | FAS, PPS | Non-<br>inferiority of<br>HDq12 vs<br>2q8 and non-<br>inferiority of<br>HDq16 vs<br>2q8 in FAS | MMRM | LOCF<br>ANCOVA:<br>MI with<br>ANCOVA,<br>tipping<br>point<br>analysis | Yes, for<br>subgroups sex,<br>age, race,<br>ethnicity,<br>geographic<br>region, baseline<br>BCVA<br>category,<br>baseline CRT<br>category, prior<br>DME treatment | Superiority<br>of HDq12<br>vs 2q8 and<br>superiority<br>of HDq16<br>vs 2q8 |
| Secondary Endpoi | nts | | | | | |
| Change from<br>baseline in BCVA<br>at Week 60 | FAS, PPS | Non-<br>inferiority of<br>HDq12 vs<br>2q8 and non-<br>inferiority of<br>HDq16 vs<br>2q8 in FAS | MMRM | Non-<br>inferiority in<br>PPS; LOCF<br>ANCOVA:<br>MI with<br>ANCOVA | Yes, for<br>subgroups sex,<br>age, race,<br>ethnicity,<br>geographic<br>region, baseline<br>BCVA<br>category,<br>baseline CRT<br>category, prior<br>DME treatment | Superiority<br>of HDq12<br>vs 2q8 and<br>superiority<br>of HDq16<br>vs 2q8 |
| Proportion of patients with a ≥2 step improvement in DRSS at week 48 | FAS | Non-<br>inferiority of<br>HDq12 vs<br>2q8 and non-<br>inferiority of<br>HDq16 vs<br>2q8 in FAS | CMH test<br>with LOCF | OC | Yes, for<br>subgroups sex,<br>age, race,<br>ethnicity,<br>geographic<br>region, baseline<br>BCVA<br>category,<br>baseline CRT<br>category, prior<br>DME treatment | No |

Protocol: VGFTe-HD-DME-1934

| Endpoint | Analysis<br>Populations | Primary<br>Analysis | Statistical<br>Method | Supportive<br>Analysis | Subgroup<br>Analysis | Other<br>Analyses |
|---|---|---|---|---|---|---|
| Proportion of patients gaining ≥ 15 letters in BCVA from baseline at week 48 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | OC | No | No |
| Proportion of patients with BCVA ≥ 69 letters at week 48 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | OC | No | No |
| Change from baseline in CRT at week 48 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | MMRM | No | No | No |
| Proportion of patients without leakage on FA at week 48 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | No | No | No |
| Change from<br>baseline in NEI-<br>VFQ total score at<br>week 48 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | MMRM | No | No | No |
| Proportion of patients without retinal fluid (total fluid, IRF, and/or SRF) at the foveal center and in center subfield at week 48, 60, and 96 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | No | No | No |
| Time to fluid-free<br>retina over 48, 60,<br>and 96 weeks<br>(total fluid, IRF<br>and/or SRF at<br>foveal center and<br>in the center<br>subfield) | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | Kaplan-<br>Meier | No | No | No |

| Endpoint | Analysis<br>Populations | Primary<br>Analysis | Statistical<br>Method | Supportive<br>Analysis | Subgroup<br>Analysis | Other<br>Analyses |
|---|---|---|---|---|---|---|
| Proportion of patients with sustained fluid-free retina over 48, 60, and 96 weeks (total fluid, IRF and/or SRF at foveal center and in the center subfield) | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | No | No | No |
| Time to sustained fluid-free retina over 48, 60, and 96 weeks (total fluid, IRF and/or SRF at foveal center and in the center subfield) | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | Kaplan-<br>Meier | No | No | No |
| Proportion of patients without CSME at week 48, 60, and 96 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | No | No | No |
| Proportion of patients with $a \ge 3$ step improvement in DRSS at week 48, 60, and 96 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | OC | No | No |
| Proportions of patients gaining and losing $\geq 5$ or $\geq 10$ letters at week 48, 60, and 96 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | OC | No | No |
| Proportion of patients losing ≥ 15 letters at week 48, 60, and 96 | FAS | HDq12 vs<br>2q8 and<br>HDq16 vs<br>2q8 | CMH test<br>with LOCF | OC | No | No |
| Proportion of patients randomized to HDq16 maintaining q16 dosing interval or longer through weeks 48, 60, and 96 | FAS | Descriptive | Descriptive statistics | No | No | No |

| Endpoint | Analysis<br>Populations | Primary<br>Analysis | Statistical<br>Method | Supportive<br>Analysis | Subgroup<br>Analysis | Other<br>Analyses |
|---|---|---|---|---|---|---|
| Proportion of patients randomized to HDq12 maintaining q12 dosing interval or longer through weeks 48, 60 and 96 | FAS | Descriptive | Descriptive statistics | No | No | No |
| Proportion of patients with an assigned injection interval of ≥16 or ≥20 weeks based on assessment at the last injection visit | FAS | Descriptive | Descriptive statistics | No | No | No |

## **Safety Analyses:**

| Endpoint | Analysis | Primary | Statistical | Supportive | Subgroup | Other |
|---|---|---|---|---|---|---|
| | Populations | Analysis | Method | Analysis | Analysis | Analyses |
| Adverse events | SAF | Percent of patients by SOC and PT: Up to Week 48 Up to Week 60 Up to Week 96 | Descriptive statistics | No | Yes, for subgroups sex, age, race, ethnicity, geographic region (Note: only for Ocular TEAEs in study eye, non-ocular TEAEs, Serious ocular TEAEs in study eye, Serious non-ocular TEAEs) Subset analysis in those patients who receive bilateral aflibercept treatment | Overall summary, ocular TEAE in study eye, ocular TEAE in fellow eye, non-ocular TEAE, drugrelated AE, injection-procedure-related TEAE, study-conduct-related TEAE, 2mg-aflibercept-in-the-fellow-eye-related TEAE, teading to discontinuation, SAEs, drugrelated SAEs, injection-procedure-related SAE, study-conduct-related SAE, study-conduct-related SAE, 2mg-aflibercept-in-the-fellow-eye-related SAE, 2mg-aflibercept-in-the-fellow-eye-related SAE, 2mg-aflibercept-in-the-fellow-eye-related SAE, 2mg-aflibercept-in-the-fellow-eye-related SAE, Deaths, APTC events, intraocular inflammation events, and nasal mucosa events |

| Endpoint | Analysis<br>Populations | Primary<br>Analysis | Statistical<br>Method | Supportive<br>Analysis | Subgroup<br>Analysis | Other<br>Analyses |
|---|---|---|---|---|---|---|
| Clinical<br>laboratory<br>measurement<br>s (chemistry,<br>hematology,<br>urinalysis,<br>HbA1c) | SAF | Summary by visit including changes from baseline | Descriptive statistics | No | No | Shift tables,<br>PCSV summary |
| Vital signs<br>(temperature,<br>pulse, and<br>blood<br>pressure) | SAF | Summary by visit including changes from baseline | Descriptive statistics | No | No | No |
| 12-Lead ECG | SAF | Summary by<br>visit including<br>changes from<br>baseline | Descriptive statistics | No | No | ECG status<br>(normal/abnorm<br>al) by visit, shift<br>tables of ECG<br>status |
| Intraocular pressure | SAF | Summary by visit including changes from baseline | Descriptive statistics | No | No | Proportions of patients with ≥ 10 mmHg increase in IOP measurement from baseline to any pre-dose measurement, > 21 mmHg for any pre-dose measurement, ≥ 25 mmHg for any pre-dose measurement, ≥ 35 mmHg at any time |
| Surgical procedures | SAF | Ocular<br>surgeries in the<br>study eye,<br>percent of<br>patients by PT | Descriptive statistics | No | No | Ocular<br>surgeries in the<br>fellow eye, non-<br>ocular surgeries |

## 10.2. Schedule of Time and Events

## 10.2.1. Schedule of Time and Events (Main study)

## **∄**Baseline to Week 48

| Dascinic to Week 40 | | 1 | 1 | | | | | | | | | | T | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Screen-<br>ing | Base-<br>line | Visit | Visit | Optional<br>Visit | Visit | Visit | Visit | Visit | Visit | Visit | Visit | Visit | Visit | Visit |
| , | Visit 1 | Visit 2 | 3 | 4 | 4.1 <sup>1</sup> | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Week | | 0 | 4 | 8 | | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 |
| Day | -21 to<br>-1 | 1 | 29 | 57 | 60-64 | 85 | 113 | 141 | 169 | 197 | 225 | 253 | 281 | 309 | 337 |
| Window (day) | | | ±5 | ±5 | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 |
| Screening/Baseline: | | | | | | | | | | | | | | | |
| Informed consent<br>form(ICF) | X | | | | | | | | | | | | | | |
| Dense PK substudy ICF <sup>2</sup> | X | | | | | | | | | | | | | | |
| Genomic substudy ICF3 | X | | | | | | | | | | | | | | |
| Future Biomedical<br>Research ICF <sup>4</sup> | X | | | | | | | | | | | | | | |
| Inclusion/Exclusion | X | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Randomization | | X | | | | | | | | | | | | | |
| Administer Study Drug <sup>5</sup> | | | | | | | | | | | | | | | |
| Study drug (active or sham) | | X | X | X | | X | X | X | X | Х | Х | X | X | X | X |
| DRM assessment | | | | | | | $X^6$ | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | $X^6$ | $X^6$ |
| Ocular Efficacy and Safe | ety (bilater | al unless in | dicated): | | | | | | | | | | | | |
| BCVA (ETDRS) and<br>Refraction <sup>7</sup> | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| IOP8 | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| Slit lamp examination | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| Indirect<br>ophthalmoscopy <sup>9</sup> | X | X | X | X | | X | X | X | X | X | X | X | X | X | x |
| FA, FP <sup>10</sup> | X | | | | | X | | | X | | | X | | | X |
| SD-OCT <sup>10</sup> | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |

## Baseline to Week 48 (continued)

| <u>'</u> | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedure | Screen-<br>ing<br>Visit 1 | Base-<br>line<br>Visit 2 | Visit<br>3 | Visit<br>4 | Optional<br>Visit<br>4.1 <sup>1</sup> | Visit<br>5 | Visit<br>6 | Visit | Visit<br>8 | Visit<br>9 | Visit<br>10 | Visit<br>11 | Visit<br>12 | Visit<br>13 | Visit<br>14 |
| Week | | 0 | 4 | 8 | | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 |
| Day | -21 to<br>-1 | 1 | 29 | 57 | 60-64 | 85 | 113 | 141 | 169 | 197 | 225 | 253 | 281 | 309 | 337 |
| Window (day) | | | ±5 | ±5 | | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 |
| OCTA substudies <sup>11</sup> | X | | | | | X | | | X | | | X | | | X |
| NEI-VFQ-25 | X | | | | | | | | X | | | | | | X |
| Nonocular Safety: | | | | | | | | | | | | | | | |
| Physical examination | X | | | | | | | | | | | | | | |
| Vital signs <sup>12</sup> | X | X | X | X | X <sup>1</sup> | X | X | X | X | X | X | X | X | X | X |
| ECG | X | | | | | | | | | | | | | | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Laboratory Testing <sup>13</sup> | | | | | | | | | | | | | | | |
| Hematology | X | | | | | | | | | | | | | | X |
| Blood chemistry | X | | | | | | | | | | | | | | X |
| HbA1c | X | | | | | | | | | | | | | | X |
| Pregnancy test (women<br>of childbearing potential) <sup>14</sup> | X<br>Serum | X<br>Urine | X<br>Urine | X<br>Urine | | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine |
| Urinalysis/UPCR | X | | | | | | | | | | | | | | X |
| Pharmacokinetics and O | ther Samp | | | | | | | | | | | | | | |
| PK samples (Dense) <sup>15, 17</sup> | | See schedule<br>below | X | | X <sup>1</sup> | X | | | | X | | | | | X |
| PK samples (Sparse) <sup>16, 17</sup> | | X | X | | $X^1$ | X | | | | X | | | | | X |
| Genomic DNA sample <sup>3</sup> | | X | | | | | | | | | | | | | |
| Immunogenicity<br>sample <sup>16, 17</sup> | | X | | | | | | | | | | | | | Х |

## **Neek 52 to Week 96**

| Study Procedure | Visit<br>15 | Visit<br>16 | Visit<br>17 | Visit<br>18 | Visit<br>19 | Visit<br>20 | Visit<br>21 | Visit<br>22 | Visit<br>23 | Visit<br>24 | Visit<br>25 | EOS<br>Visit <sup>18</sup><br>26 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | 52 | 56 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| Day | 365 | 393 | 421 | 449 | 477 | 505 | 533 | 561 | 589 | 617 | 645 | 673 |
| Window (day) | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 | ±5 |
| Screening/Baseline: | | | | | | | | | | | | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Administer Study Drug | 5 | • | • | • | • | | | | | • | • | • |
| Study Drug (active or sham) | X | X | X | X | X | X | X | X | X | X | X | |
| DRM assessment | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | X <sup>6</sup> | |
| Ocular Efficacy and Sa | fety (bilate | ral unless | indicated): | | | | • | | | | | |
| BCVA (ETDRS) and refraction <sup>7</sup> | х | Х | Х | X | Х | Х | Х | Х | X | Х | Х | Х |
| IOP8 | X | X | X | X | X | X | X | X | X | X | X | X |
| Slit lamp examination | X | X | X | X | X | X | X | X | X | X | X | X |
| Indirect ophthalmoscopy9 | х | х | Х | Х | х | Х | х | х | X | Х | Х | Х |
| FA, FP <sup>10</sup> | | | X | | | X | | | X | | | X |
| SD-OCT <sup>10</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| OCTA Substudies <sup>11</sup> | | | X | | | X | | | X | | | X |
| NEI VFQ-25 | | | X | | | | | | | | | X |
| Nonocular Safety: | | | | | | | | | | | | |
| Physical examination | | | | | | | | | | | | |
| Vital signs <sup>12</sup> | X | X | X | X | X | X | X | X | X | X | X | X |
| ECG | | | | | | | | | | | | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X |
| Laboratory Testing <sup>13</sup> | 1 | 1 | T | 1 | 1 | 1 | | ı | | | | |
| Hematology | | | | | | | | | | | | X |
| Blood chemistry | | | | | | | | | | | | X |
| HbA1c | | | | | | | | | | | | X |

| Study Procedure | Visit<br>15 | Visit<br>16 | Visit<br>17 | Visit<br>18 | Visit<br>19 | Visit<br>20 | Visit<br>21 | Visit<br>22 | Visit<br>23 | Visit<br>24 | Visit<br>25 | EOS<br>Visit <sup>18</sup><br>26 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Week | 52 | 56 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| Day | 365 | 393 | 421 | 449 | 477 | 505 | 533 | 561 | 589 | 617 | 645 | 673 |
| Pregnancy test (women<br>of childbearing<br>potential) <sup>14</sup> | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | X<br>Urine | |

Date: 19 AUGUST 2022

| Offinalysis/OPCR | Λ |
|-------------------------------------|---|
| Pharmacokinetics and Other Sampling | |
| PK samples(Dense) <sup>15,17</sup> | |
| PK samples(Sparse)16,17 | |
| Genomic DNA sample <sup>3</sup> | |
| Immunogenicity | v |
| sample <sup>16, 17</sup> | |

BCVA=Best corrected visual acuity, DRM = Dose regimen modification, ECG=electrocardiogram, ETDRS=Early Treatment Diabetic Retinopathy Study, FA=fluorescein angiography, FP=fundus photography, IOP=Intraocular pressure, OCTA = optical coherence tomography angiography, PK=pharmacokinetics, SD-OCT=spectral domain optical coherence tomography, UPCR=urine protein:creatinine ratio, UWFA = ultra-widefield fluorescein angiography.

#### Footnotes for the Schedule of Events

1. An optional visit for all patients on days 60 to 64 (after the third injection) to collect a PK sample and assess heart rate and BP (no temperature measures required) as well as concomitant medications and AEs

Protocol: VGFTe-HD-DME-1934

- 2. Signed only by patients participating in the dense PK substudy and in addition to the study ICF
- 3. The optional genomic substudy ICF should be presented to patients at the screening visit and may be signed at any subsequent visit at which the patient chooses to participate after screening. The genomic DNA sample should be collected on day 1/baseline (pre-dose) or at any study visit from patients who have signed the substudy ICF.
- 4. The optional future biomedical research substudy ICF should be presented to patients and signed at the screening visit.
- 5. Refer to pharmacy manual for study drug injection guidelines. Following study drug injection, patients will be observed for approximately 30 minutes.
- 6. Assessments for DRM criteria will occur in all patients at all visits for masking purposes beginning at week 16. Actual DRMs will be implemented as described in Section 6.1.
- 7. Patients enrolled at sites participating in the optional visual function substudy may undergo additional visual function tests. See study procedure manual for details.
- 8. Intraocular pressure will be measured at all study visits (bilateral). On days when study drug is administered, IOP should be measured pre-dose (bilaterally) by the masked investigator (or designee) and approximately 30 minutes after administration of study drug (study eye only) by the unmasked investigator (or designee). IOP will be measured using Goldmann applanation tonometry or Tono-pen<sup>TM</sup> and the same method of measurement must be used in each patient throughout the study.
- 9. Indirect ophthalmoscopy will be performed bilaterally at all visits by the masked investigator. On days when study drug is administered, it should also be performed immediately after administration of study drug (study eye only) by the unmasked investigator.
- 10. The same SD-OCT/FA/FP imaging system used at screening and day 1 must be used at all follow-up visits in each patient. Images will be taken in both eyes before dosing at each required visit. For FA, the study eye will be the transit eye and images should be collected using the widest field available. If available, sites should also submit an optional ultra-widefield color photograph.
- 11. Details on an optional substudy evaluating OCTA are provided in study procedure manual. Images will be collected at the same timepoints as FA/FP.
- 12. Vital signs (BP, heart rate, temperature) should be measured prior to injection and any blood sampling. When possible, timing of all BP assessments should be within 2 hours of clock time of dosing on day 1. Table 3 in protocol shows additional measurements for patients enrolled in the dense PK substudy.

Regeneron Pharmaceuticals, Inc. Statistical Analysis Plan

- 13. All samples collected for laboratory assessments should be obtained prior to administration of fluorescein and prior to administration of study drug.
- 14. For women of childbearing potential, a negative serum pregnancy test at screening is required for eligibility. A negative urine pregnancy test is required before treatment is administered at subsequent visits.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

- 15. Dense PK sampling will be performed in approximately 24 patients (n=8/group) as indicated in Table 2. Additional samples will be drawn according to the dense PK substudy schedule defined in Table 3 in protocol. On dosing visits, PK sampling should be performed prior to the administration of study drug and within 2 hours of the clock time of dosing on day 1.
- 16. On dosing visits, PK and ADA sampling will be performed prior to dosing.
- 17. PK and ADA samples may also be drawn at any non-specified scheduled visit or any unscheduled visit if a patient experiences an unexpected SAE.
- 18. The EOS will also represent the early termination visit.

#### 10.2.2. Schedule of Time and Events (Dense PK substudy)

| Visit | Dose | Assessment<br>Day | Assessment Time<br>(h) | PK Sample | Heart Rate and<br>Blood Pressure <sup>3</sup> |
|---|---|---|---|---|---|
| Screening 21 | | -20 to -1 | ±2h | | $X^2$ |
| | | | Predose <sup>3</sup> | X | $X^2$ |
| Visit 2 | X | 1 | 4h ±30min | X | |
| | | | 8h ±2h | X | |
| | | 2 | ±2h <sup>3</sup> | X | $X^2$ |
| | | 3 | ±2h <sup>3</sup> | X | $X^2$ |
| | | 5 | ±2h <sup>3</sup> | X | $X^2$ |
| | | <u>8</u> | ±2h <sup>3</sup> | X | $X^2$ |
| | | 15 | ±2h <sup>3</sup> | X | $X^2$ |
| | | 22 | ±2h <sup>3</sup> | X | $X^2$ |

## 10.3. NEI-VFQ-25 Sub-scale Scores and Total Score

The calculation for NEI-VFQ-25 sub-scale scores and total score will be performed according to The National Eye Institute (2000). The algorithm is then: As a preparation of the VFQ-25 calculation, the items of the questionnaire will be recoded according to Table 3. In the further calculations, only the recoded item values will be used. For the recoded values, they generally represent the best possible result as "100" and the worst possible result as "0".

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

Table 3: Recoding of NEI-VFQ 25 items

| Item no. | Original response to | Recoded item |
|---|---|---|
| 1, 3, 4, 15c <sup>(a)</sup> | 1 | 100 |
| | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| 2 | 1 | 100 |
| | 2 | 80 |
| | 3 | 60 |
| | 4 | 40 |
| | 5 | 20 |
| | 6 | 0 |
| 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 16a | 1 | 100 |
| , | 2 | 75 |
| | 3 | 50 |
| | 4 | 25 |
| | 5 | 0 |
| | 6 | * |
| 17, 18, 19, 20, 21, 22, 23, 24, 25 | 1 | 0 |
| , -, -, -, , , -, , - | 2 | 25 |
| | 3 | 50 |
| | 4 | 75 |
| | 5 | 100 |

<sup>(</sup>a) Item 15c has four-response levels but is expanded to a five-levels using item 15b: if 15b="1", then 15c="0" / if 15b=("2" or "3"), then 15c="missing"

For the VFQ questionnaire, 12 sub-scal. es will be evaluated (see Table 4), and 11 of these sub-scales will be included in the total VFQ score.

<sup>\*</sup> Here, Response choice "6" indicates that the person does not perform the activity because of non-vision-related problems. If this choice is selected, the item is coded as "missing".

Table 4: Sub-scales of the NEI-VFQ 25 score

| Sub-scale no. | Sub-scale | | Number of items | (Recoded)<br>items to be<br>averaged | Sub-scale included in total scale |
|---|---|---|---|---|---|
| 1 | General Health | 1 | | 1 | No |
| 2 | General Vision | 1 | | 2 | Yes |
| 3 | Ocular Pain | 2 | | 4, 19 | Yes |
| 4 | Near Activities | 3 | | 5, 6, 7 | Yes |
| 5 | Distance Activities Vision specific: | 3 | | 8, 9, 14 | Yes |
| 6 | Social Functionin | g2 | | 11, 13 | Yes |
| 7 | Mental Health | 4 | | 3, 21, 22, 25 | Yes |
| 8 | Role Difficulties | 2 | | 17, 18 | Yes |
| 9 | Dependency | 3 | | 20, 23, 24 | Yes |
| 10 | Driving | 3 | | 15c, 16, 16a | Yes |
| 11 | Color vision | 1 | | 12 | Yes |
| 12 | Peripheral Vision | 1 | | 10 | Yes |

Date: 19 AUGUST 2022

For a single sub-scale, the value will be determined as the average of the non-missing recoded item values assigned to this sub-scale. A sub-scale value will only be assessed as missing if all items for this sub-scale have "missing" as a result.

The total score is calculated as the arithmetic mean of all non-missing sub-scales (except General Health):

$$total\ result = \frac{(sum\ of\ non\ - missing\ sub\ -\ scale\ values)}{Total\ number\ of\ sub\ -\ scales\ with\ non\ - missing\ result}$$

Due to this calculation approach, the total result will be non-missing if at least one sub-scale result is non-missing.

# 10.4. Detailed Definitions of Special AE Categories and Medical History Subgroups

Prior to database lock these preferred terms will be updated as necessary based on the current MedDRA version.

#### 10.4.1. Medical history and AE grouping of hypertension

| Preferred term |
|----------------------------------------|
| Accelerated hypertension |
| Blood pressure ambulatory increased |
| Blood pressure diastolic increased |
| Blood pressure inadequately controlled |
| Blood pressure increased |
| Blood pressure systolic increased |

Regeneron Pharmaceuticals, Inc. Statistical Analysis Plan

| Preferred term |
|----------------------------------------|
| Diastolic hypertension |
| Endocrine hypertension |
| Essential hypertension |
| Hypertension |
| Hypertension neonatal |
| Hypertensive angiopathy |
| Hypertensive cardiomegaly |
| Hypertensive cardiomyopathy |
| Hypertensive cerebrovascular disease |
| Hypertensive crisis |
| Hypertensive emergency |
| Hypertensive encephalopathy |
| Hypertensive end-organ damage |
| Hypertensive heart disease |
| Hypertensive nephropathy |
| Hypertensive urgency |
| Labile hypertension |
| Malignant hypertension |
| Malignant hypertensive heart disease |
| Malignant renal hypertension |
| Maternal hypertension affecting foetus |
| Mean arterial pressure increased |
| Neurogenic hypertension |
| Orthostatic hypertension |
| Page kidney |
| Prehypertension |
| Renal hypertension |
| Renovascular hypertension |
| Retinopathy hypertensive |
| Supine hypertension |
| Systolic hypertension |
| White coat hypertension |

Protocol: VGFTe-HD-DME-1934

## 10.4.2. AE grouping of intraocular inflammation

| Preferred term |
|--------------------------------|
| Anterior chamber cell |
| Anterior chamber fibrin |
| Anterior chamber flare |
| Anterior chamber inflammation |
| Aqueous fibrin |
| Autoimmune uveitis |
| Candida endophthalmitis |
| Chorioretinitis |
| Choroiditis |
| Cyclitis |
| Endophthalmitis |
| Eye infection |
| Eye infection bacterial |
| Eye infection chlamydial |
| Eye infection fungal |
| Eye infection intraocular |
| Eye infection staphylococcal |
| Eye inflammation |
| Нуроруоп |
| Infectious iridocyclitis |
| Infective iritis |
| Infective uveitis |
| Iridocyclitis |
| Iritis |
| Mycotic endophthalmitis |
| Necrotising retinitis |
| Non-infectious endophthalmitis |
| Noninfective chorioretinitis |
| Pseudoendophthalmitis |
| Uveitis |
| Vitreal cells |
| Vitreous fibrin |
| Vitritis |

Protocol: VGFTe-HD-DME-1934

## 10.4.3. AE grouping of nasal mucosal events

| Preferred term |
|-----------------------|
| Epistaxis |
| Nasal inflammation |
| Nasal mucosal erosion |
| Nasal mucosal ulcer |
| Nasal ulcer |

#### 10.4.4. Medical history of renal impairment

Renal impairment is defined by CRCL values.

Categories for renal impairment:

- CLCR >80ml/min (normal),
- CLCR >50-80ml/min (mild),
- CLCR >30-50 ml/min (moderate),
- CLCR <=30ml/min or 'requiring dialysis' (severe)

CLCR will be calculated using baseline values (creatinine, age, weight, sex) using the Cockcroft-Gault equation:

Males: CLCR = (140-age)\*body weight / (72\*creatinine in mg/dL)

Females: CLCR = (140-age)\*body weight\*0.85 / (72\*creatinine in mg/dL)

#### 'Requiring dialysis' is defined by PT in medical history

| Preferred Term |
|-------------------------------|
| Continuous haemodiafiltration |
| Dialysis |
| Dialysis device insertion |
| Haemodialysis |
| Haemofiltration |
| Peritoneal dialysis |
| Removal of renal transplant |
| Renal replacement therapy |
| Renal transplant |

Protocol: VGFTe-HD-DME-1934

## 10.4.5. Medical history of hepatic impairment

| Preferred term |
|---------------------------------------------|
| 5'nucleotidase increased |
| AST to platelet ratio index increased |
| AST/ALT ratio abnormal |
| Accessory liver lobe |
| Acquired antithrombin III deficiency |
| Acquired factor IX deficiency |
| Acquired factor V deficiency |
| Acquired factor VIII deficiency |
| Acquired factor XI deficiency |
| Acquired hepatocerebral degeneration |
| Acquired protein S deficiency |
| Acute graft versus host disease in liver |
| Acute hepatic failure |
| Acute hepatitis B |
| Acute hepatitis C |
| Acute on chronic liver failure |
| Acute yellow liver atrophy |
| Adenoviral hepatitis |
| Alagille syndrome |
| Alanine aminotransferase abnormal |
| Alanine aminotransferase increased |
| Alcoholic encephalopathy |
| Alcoholic liver disease |
| Allergic hepatitis |
| Alloimmune hepatitis |
| Ammonia abnormal |
| Ammonia increased |
| Anorectal varices |
| Anorectal varices haemorrhage |
| Anti factor X activity abnormal |
| Anti factor X activity decreased |
| Anti factor X activity increased |
| Anti-liver cytosol antibody type 1 positive |
| Antithrombin III decreased |
| Ascites |
| Aspartate aminotransferase abnormal |
| Aspartate aminotransferase increased |
| Asterixis |
| Asymptomatic viral hepatitis |
| Autoimmune hepatitis |

Protocol: VGFTe-HD-DME-1934

| Preferred term |
|--------------------------------------------|
| Bacterascites |
| Benign hepatic neoplasm |
| Benign hepatobiliary neoplasm |
| Benign recurrent intrahepatic cholestasis |
| Bile output abnormal |
| Bile output decreased |
| Biliary ascites |
| Biliary cirrhosis |
| Biliary fibrosis |
| Bilirubin conjugated abnormal |
| Bilirubin conjugated increased |
| Bilirubin excretion disorder |
| Bilirubin urine present |
| Biopsy liver abnormal |
| Blood alkaline phosphatase abnormal |
| Blood alkaline phosphatase increased |
| Blood bilirubin abnormal |
| Blood bilirubin increased |
| Blood bilirubin unconjugated increased |
| Blood cholinesterase abnormal |
| Blood cholinesterase decreased |
| Blood fibrinogen abnormal |
| Blood fibrinogen decreased |
| Blood thrombin abnormal |
| Blood thrombin decreased |
| Blood thromboplastin abnormal |
| Blood thromboplastin decreased |
| Bromosulphthalein test abnormal |
| Cardiohepatic syndrome |
| Cerebrohepatorenal syndrome |
| Child-Pugh-Turcotte score abnormal |
| Child-Pugh-Turcotte score increased |
| Cholaemia |
| Cholangiosarcoma |
| Cholestasis |
| Cholestatic liver injury |
| Cholestatic pruritus |
| Chronic graft versus host disease in liver |
| Chronic hepatic failure |
| Chronic hepatitis |
| Chronic hepatitis B |

| Preferred term |
|-----------------------------------------------|
| Chronic hepatitis C |
| Cirrhosis alcoholic |
| Coagulation factor IX level abnormal |
| Coagulation factor IX level decreased |
| Coagulation factor V level abnormal |
| Coagulation factor V level decreased |
| Coagulation factor VII level abnormal |
| Coagulation factor VII level decreased |
| Coagulation factor X level abnormal |
| <u> </u> |
| Coagulation factor X level decreased |
| Coagulation factor decreased |
| Coma hepatic |
| Complications of transplanted liver |
| Computerised tomogram liver abnormal |
| Congenital absence of bile ducts |
| Congenital hepatic fibrosis |
| Congenital hepatitis B infection |
| Congenital hepatitis C infection |
| Congenital hepatobiliary anomaly |
| Congenital hepatomegaly |
| Congenital viral hepatitis |
| Congestive hepatopathy |
| Cryptogenic cirrhosis |
| Cystic fibrosis hepatic disease |
| Cytokeratin 18 increased |
| Cytomegalovirus hepatitis |
| Deficiency of bile secretion |
| Diabetic hepatopathy |
| Dilatation intrahepatic duct congenital |
| Drug-induced liver injury |
| Duodenal varices |
| Fatty liver alcoholic |
| Flood syndrome |
| Focal nodular hyperplasia |
| Foetor hepaticus |
| Galactose elimination capacity test abnormal |
| Galactose elimination capacity test decreased |
| Gallbladder varices |
| Gamma-glutamyltransferase abnormal |
| Gamma-glutamyltransferase increased |
| Gastric variceal injection |

| Preferred term |
|---------------------------------------------------|
| Gastric variceal ligation |
| Gastric varices Gastric varices |
| Gastric varices Gastric varices haemorrhage |
| Gastroesophageal variceal haemorrhage prophylaxis |
| Gianotti-Crosti syndrome |
| Glutamate dehydrogenase increased |
| Glycocholic acid increased |
| Glycogen storage disease type I |
| Glycogen storage disease type III |
| , |
| Glycogen storage disease type IV |
| Glycogen storage disease type VI |
| Graft versus host disease in liver |
| Granulomatous liver disease |
| Guanase increased |
| HBV-DNA polymerase increased |
| Haemangioma of liver |
| Haemorrhagic ascites |
| Haemorrhagic hepatic cyst |
| Hepaplastin abnormal |
| Hepaplastin decreased |
| Hepatectomy |
| Hepatic adenoma |
| Hepatic amoebiasis |
| Hepatic angiosarcoma |
| Hepatic artery flow decreased |
| Hepatic atrophy |
| Hepatic calcification |
| Hepatic cancer |
| Hepatic cancer metastatic |
| Hepatic cancer recurrent |
| Hepatic cancer stage I |
| Hepatic cancer stage II |
| Hepatic cancer stage III |
| Hepatic cancer stage IV |
| Hepatic candidiasis |
| Hepatic cirrhosis |
| Hepatic cyst |
| Hepatic cyst infection |
| Hepatic cyst ruptured |
| Hepatic cytolysis |
| Hepatic echinococciasis |

| Preferred term |
|--------------------------------------------------------------|
| Hepatic encephalopathy |
| Hepatic encephalopathy prophylaxis |
| Hepatic enzyme abnormal |
| Hepatic enzyme decreased |
| Hepatic enzyme increased |
| Hepatic failure |
| Hepatic fibrosis |
| Hepatic fibrosis marker abnormal |
| Hepatic fibrosis marker increased |
| Hepatic function abnormal |
| Hepatic gas gangrene |
| Hepatic haemangioma rupture |
| Hepatic hamartoma |
| Hepatic hydrothorax |
| Hepatic hypertrophy |
| Hepatic hypoperfusion |
| Hepatic infection |
| Hepatic infection bacterial |
| Hepatic infection fungal |
| Hepatic infection helminthic |
| Hepatic infiltration eosinophilic |
| Hepatic lesion |
| Hepatic lipoma |
| Hepatic lymphocytic infiltration |
| Hepatic mass |
| Hepatic necrosis |
| Hepatic neoplasm |
| Hepatic neuroendocrine tumour |
| Hepatic pain |
| Hepatic perfusion disorder |
| Hepatic sarcoma |
| Hepatic sequestration |
| Hepatic steato-fibrosis |
| Hepatic steatosis |
| Hepatic vascular resistance increased |
| Hepatic venous pressure gradient abnormal |
| Hepatic venous pressure gradient increased |
| Hepatitis |
| Hepatitis A |
| Hepatitis A antibody abnormal |
| Hepatitis A antibody positive Hepatitis A antibody positive |
| Tiepanus A annoug positive |

| Dueformed town |
|---------------------------------------|
| Preferred term |
| Hepatitis A antigen positive |
| Hepatitis A immunity confirmed |
| Hepatitis A virus test positive |
| Hepatitis B |
| Hepatitis B DNA assay positive |
| Hepatitis B DNA increased |
| Hepatitis B antibody abnormal |
| Hepatitis B antibody positive |
| Hepatitis B antigen positive |
| Hepatitis B core antibody positive |
| Hepatitis B core antigen positive |
| Hepatitis B e antibody positive |
| Hepatitis B e antigen positive |
| Hepatitis B immunity confirmed |
| Hepatitis B reactivation |
| Hepatitis B surface antibody positive |
| Hepatitis B surface antigen positive |
| Hepatitis B virus test positive |
| Hepatitis C |
| Hepatitis C RNA increased |
| Hepatitis C RNA positive |
| Hepatitis C antibody positive |
| Hepatitis C core antibody positive |
| Hepatitis C virus test positive |
| Hepatitis D |
| Hepatitis D RNA positive |
| Hepatitis D antibody positive |
| Hepatitis D antigen positive |
| Hepatitis D virus test positive |
| Hepatitis E |
| Hepatitis E RNA positive |
| Hepatitis E antibody abnormal |
| Hepatitis E antibody positive |
| Hepatitis E antigen positive |
| Hepatitis E immunity confirmed |
| Hepatitis E virus test positive |
| Hepatitis F |
| Hepatitis G |
| Hepatitis H |
| Hepatitis acute |
| Hepatitis alcoholic |

| Preferred term |
|--------------------------------------|
| Hepatitis cholestatic |
| Hepatitis chronic active |
| Hepatitis chronic persistent |
| Hepatitis fulminant |
| Hepatitis infectious mononucleosis |
| Hepatitis mumps |
| Hepatitis neonatal |
| Hepatitis non-A non-B |
| Hepatitis non-A non-B non-C |
| Hepatitis post transfusion |
| Hepatitis syphilitic Hepatitis toxic |
| Hepatitis toxoplasmal |
| Hepatitis viral |
| Hepatitis viral test positive |
| Hepato-lenticular degeneration |
| Hepatobiliary cancer |
| Hepatobiliary cancer in situ |
| Hepatobiliary cyst |
| Hepatobiliary disease |
| Hepatobiliary infection |
| Hepatobiliary neoplasm |
| Hepatobiliary scan abnormal |
| Hepatoblastoma |
| Hepatoblastoma recurrent |
| Hepatocellular carcinoma |
| Hepatocellular damage neonatal |
| Hepatocellular foamy cell syndrome |
| Hepatocellular injury |
| Hepatomegaly |
| Hepatopulmonary syndrome |
| Hepatorenal failure |
| Hepatorenal syndrome |
| Hepatosplenic abscess |
| Hepatosplenic candidiasis |
| Hepatosplenomegaly |
| Hepatosplenomegaly neonatal |
| Hepatotoxicity |
| Hereditary haemochromatosis |
| Herpes simplex hepatitis |
| Hyperammonaemia |

| Preferred term |
|--------------------------------------------|
| Hyperbilirubinaemia |
| Hyperbilirubinaemia neonatal |
| Hypercholia |
| Hyperfibrinolysis |
| Hypertransaminasaemia |
| Hypoalbuminaemia |
| Hypocoagulable state |
| Hypofibrinogenaemia |
| Hypoprothrombinaemia |
| Hypothrombinaemia |
| Hypothromboplastinaemia |
| Icterus index increased |
| Immune-mediated cholangitis |
| Immune-mediated hepatic disorder |
| Immune-mediated hepatitis |
| Increased liver stiffness |
| International normalised ratio abnormal |
| International normalised ratio increased |
| Intestinal varices |
| Intestinal varices haemorrhage |
| Intrahepatic portal hepatic venous fistula |
| Ischaemic hepatitis |
| Jaundice |
| Jaundice cholestatic |
| Jaundice hepatocellular |
| Jaundice neonatal |
| Kayser-Fleischer ring |
| Kernicterus |
| Leucine aminopeptidase increased |
| Liver abscess |
| Liver and pancreas transplant rejection |
| Liver carcinoma ruptured |
| Liver dialysis |
| Liver disorder |
| Liver function test abnormal |
| Liver function test decreased |
| Liver function test increased |
| Liver induration |
| Liver injury |
| Liver iron concentration abnormal |
| Liver iron concentration increased |

| Preferred term |
|------------------------------------------------------------|
| Liver opacity |
| Liver operation |
| Liver palpable |
| Liver sarcoidosis |
| Liver scan abnormal |
| Liver tenderness |
| Liver transplant |
| Liver transplant failure |
| Liver transplant rejection |
| Liver-kidney microsomal antibody positive |
| Lupoid hepatic cirrhosis |
| Lupus hepatitis |
| Magnetic resonance imaging hepatobiliary abnormal |
| Magnetic resonance proton density fat fraction measurement |
| Mitochondrial aspartate aminotransferase increased |
| Mixed hepatocellular cholangiocarcinoma |
| Mixed liver injury |
| Model for end stage liver disease score abnormal |
| Model for end stage liver disease score increased |
| Molar ratio of total branched-chain amino acid to tyrosine |
| Multivisceral transplantation |
| Necrolytic acral erythema |
| Neonatal cholestasis |
| Neonatal hepatomegaly |
| Nodular regenerative hyperplasia |
| Non-alcoholic fatty liver |
| Non-alcoholic steatohepatitis |
| Non-cirrhotic portal hypertension |
| Ocular icterus |
| Oedema due to hepatic disease |
| Oesophageal varices haemorrhage |
| Omental oedema |
| Osteopontin increased |
| Parenteral nutrition associated liver disease |
| Perihepatic discomfort |
| Perinatal HBV infection |
| Peripancreatic varices |
| Periportal oedema |
| Peritoneal fluid protein abnormal |
| Peritoneal fluid protein decreased |
| Peritoneal fluid protein increased |
| <u> </u> |
| Preferred term |
|-----------------------------------------------|
| Peritoneovenous shunt |
| Pneumobilia |
| Polycystic liver disease |
| Porphyria acute |
| Porphyria non-acute |
| Portal fibrosis |
| Portal hypertension |
| Portal hypertensive colopathy |
| Portal hypertensive enteropathy |
| Portal hypertensive gastropathy |
| Portal pyaemia |
| Portal shunt |
| Portal shunt procedure |
| Portal tract inflammation |
| Portal vein cavernous transformation |
| Portal vein dilatation |
| Portal vein flow decreased |
| Portal vein pressure increased |
| Portal venous system anomaly |
| Portopulmonary hypertension |
| Primary biliary cholangitis |
| Progressive familial intrahepatic cholestasis |
| Protein C decreased |
| Protein S abnormal |
| Protein S decreased |
| Prothrombin level abnormal |
| Prothrombin level decreased |
| Prothrombin time abnormal |
| Prothrombin time prolonged |
| Prothrombin time ratio abnormal |
| Prothrombin time ratio increased |
| Radiation hepatitis |
| Regenerative siderotic hepatic nodule |
| Renal and liver transplant |
| Retinol binding protein decreased |
| Retrograde portal vein flow |
| Reye's syndrome |
| Reynold's syndrome |
| Schistosomiasis liver |
| Small-for-size liver syndrome |
| Spider naevus |

| Preferred term |
|-----------------------------------------------------|
| Splenic artery embolisation |
| Splenic varices |
| Splenic varices haemorrhage |
| Splenorenal shunt |
| Splenorenal shunt procedure |
| Spontaneous bacterial peritonitis |
| Spontaneous intrahepatic portosystemic venous shunt |
| Steatohepatitis |
| Stomal varices |
| Subacute hepatic failure |
| Sugiura procedure |
| Sustained viral response |
| Thrombin time abnormal |
| Thrombin time prolonged |
| Total bile acids increased |
| Transaminases abnormal |
| Transaminases increased |
| Ultrasound liver abnormal |
| Urine bilirubin increased |
| Urobilinogen urine decreased |
| Urobilinogen urine increased |
| Varices oesophageal |
| Varicose veins of abdominal wall |
| Viral hepatitis carrier |
| Weil's disease |
| White nipple sign |
| Withdrawal hepatitis |
| X-ray hepatobiliary abnormal |
| Yellow skin |
| Zieve syndrome |

# 10.4.6. Medical history of cerebrovascular disease

| Agnosia Amaurosis fugax Amyloid related imaging abnormalities Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits Amyloid related imaging abnormality-oedema/effusion Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery perforation Basilar artery thrombosis |
|---|
| Amyloid related imaging abnormalities Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits Amyloid related imaging abnormality-oedema/effusion Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery perforation Basilar artery stenosis |
| Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits Amyloid related imaging abnormality-oedema/effusion Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery perforation Basilar artery stenosis |
| Amyloid related imaging abnormality-oedema/effusion Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery perforation Basilar artery stenosis |
| Amyloid related imaging abnormality-oedema/effusion Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Angiogram cerebral abnormal Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Aphasia Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Balint's syndrome Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basal ganglia haematoma Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basal ganglia haemorrhage Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basal ganglia infarction Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basal ganglia stroke Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basilar artery aneurysm Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basilar artery occlusion Basilar artery perforation Basilar artery stenosis |
| Basilar artery stenosis |
| · |
| Basilar artery thrombosis |
| Benedikt's syndrome |
| Blood brain barrier defect |
| Brachiocephalic arteriosclerosis |
| Brachiocephalic artery occlusion |
| Brachiocephalic artery stenosis |
| Brain hypoxia |
| Brain injury |
| Brain stem embolism |
| Brain stem haematoma |
| Brain stem haemorrhage |
| Brain stem infarction |
| Brain stem ischaemia |
| Brain stem microhaemorrhage |
| Brain stem stroke |
| Brain stem thrombosis |
| Brain stent insertion |
| CADASIL |
| CARASIL syndrome |
| CSF bilirubin positive |
| CSF red blood cell count positive |
| Capsular warning syndrome |
| Carotid aneurysm rupture |

Protocol: VGFTe-HD-DME-1934

| Preferred term |
|--------------------------------------------------|
| Carotid angioplasty |
| Carotid arterial embolus |
| Carotid arteriosclerosis |
| Carotid artery aneurysm |
| Carotid artery bypass |
| Carotid artery disease |
| Carotid artery dissection |
| Carotid artery dolichoectasia |
| Carotid artery insufficiency |
| Carotid artery occlusion |
| Carotid artery perforation |
| Carotid artery restenosis |
| Carotid artery stenosis |
| Carotid artery stent insertion |
| Carotid artery stent removal |
| Carotid artery thrombosis |
| Carotid endarterectomy |
| Carotid revascularisation |
| Central nervous system haemorrhage |
| Central nervous system vasculitis |
| Central pain syndrome |
| Cerebellar artery occlusion |
| Cerebellar artery thrombosis |
| Cerebellar atherosclerosis |
| Cerebellar embolism |
| Cerebellar haematoma |
| Cerebellar haemorrhage |
| Cerebellar infarction |
| Cerebellar ischaemia |
| Cerebellar microhaemorrhage |
| Cerebellar stroke |
| Cerebral amyloid angiopathy |
| Cerebral aneurysm perforation |
| Cerebral aneurysm ruptured syphilitic |
| Cerebral arteriosclerosis |
| Cerebral arteriovenous malformation haemorrhagic |
| Cerebral arteritis |
| Cerebral artery embolism |
| Cerebral artery occlusion |
| Cerebral artery perforation |
| Cerebral artery restenosis |
| Cerebral artery stenosis |

| Preferred term |
|--------------------------------------------|
| Cerebral artery stent insertion |
| Cerebral artery thrombosis |
| Cerebral capillary telangiectasia |
| Cerebral cavernous malformation |
| Cerebral circulatory failure |
| Cerebral congestion |
| Cerebral cyst haemorrhage |
| Cerebral endovascular aneurysm repair |
| Cerebral gas embolism |
| Cerebral haematoma |
| Cerebral haemorrhage |
| Cerebral haemorrhage foetal |
| Cerebral haemorrhage neonatal |
| Cerebral haemosiderin deposition |
| Cerebral hypoperfusion |
| Cerebral infarction |
| Cerebral infarction foetal |
| Cerebral ischaemia |
| Cerebral microangiopathy |
| Cerebral microembolism |
| Cerebral microhaemorrhage |
| Cerebral microinfarction |
| Cerebral reperfusion injury |
| Cerebral revascularisation |
| Cerebral septic infarct |
| Cerebral small vessel ischaemic disease |
| Cerebral thrombosis |
| Cerebral vascular occlusion |
| Cerebral vasoconstriction |
| Cerebral venous sinus thrombosis |
| Cerebral venous thrombosis |
| Cerebral ventricular rupture |
| Cerebrovascular accident |
| Cerebrovascular accident prophylaxis |
| Cerebrovascular arteriovenous malformation |
| Cerebrovascular disorder |
| Cerebrovascular insufficiency |
| Cerebrovascular pseudoaneurysm |
| Cerebrovascular stenosis |
| Charcot-Bouchard microaneurysms |
| Chronic cerebrospinal venous insufficiency |
| Claude's syndrome |

| Preferred term |
|----------------------------------------|
| Congenital cerebrovascular anomaly |
| Congenital hemiparesis |
| Delayed ischaemic neurological deficit |
| Diplegia |
| Dural arteriovenous fistula |
| Dysarthria |
| Embolic cerebellar infarction |
| Embolic cerebral infarction |
| Embolic stroke |
| Epidural haemorrhage |
| Extra-axial haemorrhage |
| Extradural haematoma |
| Extradural haematoma evacuation |
| Extraischaemic cerebral haematoma |
| Foetal cerebrovascular disorder |
| Foville syndrome |
| Haemorrhage intracranial |
| Haemorrhagic cerebellar infarction |
| Haemorrhagic cerebral infarction |
| Haemorrhagic stroke |
| Haemorrhagic transformation stroke |
| Heidelberg classification |
| Hemianaesthesia |
| Hemiasomatognosia |
| Hemiataxia |
| Hemidysaesthesia |
| Hemihyperaesthesia |
| Hemihypoaesthesia |
| Hemiparaesthesia |
| Hemiparesis |
| Hemiplegia |
| Hunt and Hess scale |
| Hypertensive cerebrovascular disease |
| Hypoxic-ischaemic encephalopathy |
| Inner ear infarction |
| Internal capsule infarction |
| Internal carotid artery deformity |
| Intra-cerebral aneurysm operation |
| Intracerebral haematoma evacuation |
| Intracranial aneurysm |
| Intracranial artery dissection |
| Intracranial haematoma |

| Preferred term |
|-------------------------------------------|
| Intracranial haemorrhage neonatal |
| Intracranial tumour haemorrhage |
| Intraventricular haemorrhage |
| Intraventricular haemorrhage neonatal |
| Ischaemic cerebral infarction |
| Ischaemic stroke |
| Lacunar infarction |
| Lacunar stroke |
| Lateral medullary syndrome |
| Lateropulsion |
| Malignant middle cerebral artery syndrome |
| Medullary compression syndrome |
| Meningorrhagia |
| Metabolic stroke |
| Migrainous infarction |
| Millard-Gubler syndrome |
| Modified Rankin score decreased |
| Modified Rankin score increased |
| Monoparesis |
| Monoplegia |
| Moyamoya disease |
| NIH stroke scale abnormal |
| NIH stroke scale score decreased |
| NIH stroke scale score increased |
| Paralysis |
| Paraparesis |
| Paraplegia |
| Paresis |
| Perinatal stroke |
| Periventricular haemorrhage neonatal |
| Pituitary apoplexy |
| Pituitary haemorrhage |
| Post cardiac arrest syndrome |
| Post procedural stroke |
| Post stroke depression |
| Posthaemorrhagic hydrocephalus |
| Precerebral arteriosclerosis |
| Precerebral artery aneurysm |
| Precerebral artery dissection |
| Precerebral artery embolism |
| Precerebral artery occlusion |
| Precerebral artery thrombosis |
| · |

| Primary familial brain calcification Pseudo-occlusion of internal carotid artery |
|---|
| Putamen haemorrhage |
| Quadriparesis |
| Quadriplegia |
| Reversible cerebral vasoconstriction syndrome |
| Reversible ischaemic neurological deficit |
| Right hemisphere deficit syndrome |
| Ruptured cerebral aneurysm |
| Septic cerebral embolism |
| Sigmoid sinus thrombosis |
| Sneddon's syndrome |
| Spinal artery embolism |
| Spinal artery thrombosis |
| Spinal cord haematoma |
| Spinal cord haemorrhage |
| Spinal cord infarction |
| Spinal cord ischaemia |
| Spinal epidural haematoma |
| Spinal epidural haemorrhage |
| Spinal stroke |
| Spinal subarachnoid haemorrhage |
| Spinal subdural haematoma |
| Spinal subdural haemorrhage |
| Spinal vascular disorder |
| Spinal vessel congenital anomaly |
| Stroke in evolution |
| Subarachnoid haematoma |
| Subarachnoid haemorrhage |
| Subarachnoid haemorrhage neonatal |
| Subclavian steal syndrome |
| Subdural haematoma |
| Subdural haematoma evacuation |
| Subdural haemorrhage |
| Subdural haemorrhage neonatal |
| Superficial siderosis of central nervous system |
| Superior sagittal sinus thrombosis |
| Susac's syndrome |
| Thalamic infarction |
| Thalamus haemorrhage |
| Thrombotic cerebral infarction |
| Thrombotic stroke |

| Preferred term |
|---------------------------------------|
| Transient ischaemic attack |
| Transverse sinus thrombosis |
| Vascular encephalopathy |
| Vascular stent occlusion |
| Vascular stent stenosis |
| Vein of Galen aneurysmal malformation |
| Vertebral artery aneurysm |
| Vertebral artery arteriosclerosis |
| Vertebral artery dissection |
| Vertebral artery occlusion |
| Vertebral artery perforation |
| Vertebral artery stenosis |
| Vertebral artery thrombosis |
| Vertebrobasilar dolichoectasia |
| Vertebrobasilar insufficiency |
| Vertebrobasilar stroke |
| Visual agnosia |
| Visual midline shift syndrome |
| Weber's syndrome |

# 10.4.7. Medical history of ischemic heart disease

| Preferred term |
|------------------------------------------------|
| Acute coronary syndrome |
| Acute myocardial infarction |
| Angina pectoris |
| Angina unstable |
| Anginal equivalent |
| Arterial revascularisation |
| Arteriogram coronary abnormal |
| Arteriosclerosis coronary artery |
| Arteriospasm coronary |
| Cardiac perfusion defect |
| Cardiac ventricular scarring |
| Chronic coronary syndrome |
| Computerised tomogram coronary artery abnormal |
| Coronary angioplasty |
| Coronary arterial stent insertion |
| Coronary artery bypass |
| Coronary artery compression |
| Coronary artery disease |
| Coronary artery dissection |
| Coronary artery embolism |
| Coronary artery insufficiency |
| Coronary artery occlusion |
| Coronary artery reocclusion |
| Coronary artery restenosis |
| Coronary artery stenosis |
| Coronary artery surgery |
| Coronary artery thrombosis |
| Coronary brachytherapy |
| Coronary bypass stenosis |
| Coronary bypass thrombosis |
| Coronary endarterectomy |
| Coronary no-reflow phenomenon |
| Coronary ostial stenosis |
| Coronary revascularisation |
| Coronary steal syndrome |
| Coronary vascular graft occlusion |
| Coronary vascular graft stenosis |
| ECG electrically inactive area |
| ECG signs of myocardial infarction |
| ECG signs of myocardial ischaemia |

Protocol: VGFTe-HD-DME-1934

| Preferred term |
|---------------------------------------------|
| Electrocardiogram PR segment depression |
| Electrocardiogram PR segment elevation |
| Electrocardiogram ST segment abnormal |
| Electrocardiogram ST segment depression |
| Electrocardiogram ST segment elevation |
| Electrocardiogram ST-T segment abnormal |
| Electrocardiogram ST-T segment depression |
| Electrocardiogram ST-T segment elevation |
| External counterpulsation |
| Haemorrhage coronary artery |
| Infarction |
| Ischaemic cardiomyopathy |
| Ischaemic contracture of the left ventricle |
| Kounis syndrome |
| Myocardial hypoperfusion |
| Myocardial hypoxia |
| Myocardial infarction |
| Myocardial ischaemia |
| Myocardial necrosis |
| Myocardial reperfusion injury |
| Myocardial stunning |
| Papillary muscle infarction |
| Percutaneous coronary intervention |
| Periprocedural myocardial infarction |
| Positive vessel remodelling |
| Post angioplasty restenosis |
| Post procedural myocardial infarction |
| Postinfarction angina |
| Prinzmetal angina |
| Scan myocardial perfusion abnormal |
| Silent myocardial infarction |
| Stent patency maintenance |
| Stress cardiomyopathy |
| Subclavian coronary steal syndrome |
| Subendocardial ischaemia |
| Vascular device occlusion |
| Vascular graft occlusion |
| Vascular graft restenosis |
| Vascular graft stenosis |
| Vascular graft thrombosis |
| Vascular stent occlusion |
| Vascular stent stenosis |

| Preferred term |
|----------------------------------|
| Ventricular compliance decreased |
| Wellens' syndrome |

# 10.5. Criteria for Potentially Clinically Significant Values (PCSV)

Protocol: VGFTe-HD-DME-1934

**Table 5: Criteria for Potentially Clinically Significant Values** 

| Parameter | Potentially clinically significant value (PCSV) |
|---|---|
| Clinical Chemistry | |
| ALT | > 3 ULN |
| AST | > 3 ULN |
| Alkaline Phosphatase | > 1.5 ULN |
| Total Bilirubin | > 1.5 ULN |
| Conjugated Bilirubin | > 35% Total Bilirubin (when Total Bilirubin >1.5 ULN) |
| ALT and Total Bilirubin | ALT > 3 ULN and Total Bilirubin > 2 ULN |
| СРК | > 3 ULN |
| Creatinine | ≥ 150 µmol/L (Adults)<br>≥ 30% from baseline |
| Uric Acid | Hyperuricemia: >408 μmol/L<br>Hypouricemia: <120 μmol/L |
| Blood Urea Nitrogen | ≥ 17 mmol/L |
| Chloride | < 80 mmol/L<br>> 115 mmol/L |
| Sodium | ≤ 129 mmol/L<br>≥ 160 mmol/L |
| Potassium | < 3 mmol/L<br>≥ 5.5 mmol/L |
| Total Cholesterol | ≥ 7.74 mmol/L (3 g/L) |
| Triglycerides | ≥ 4.6 mmol/L (4 g/L) |
| Glucose - Hypoglycaemia - Hyperglycaemia | $\leq$ 3.9 mmol/L and $\leq$ LLN $\geq$ 11.1 mmol/L (unfasted), $\geq$ 7 mmol/L (fasted) |
| HbA1c | > 8 % |
| Albumin | ≤ 25 g/L |
| Hematology | |
| WBC | < 3.0 GIGA/L (non-Black), < 2.0 GIGA/L (Black), ≥ 16.0 GIGA/L |
| Lymphocytes | > 4.0 GIGA/L |

| Parameter | Potentially clinically significant value (PCSV) |
|---|---|
| Neutrophils | < 1.5 GIGA/L (non-Black)<br>< 1.0 GIGA/L (Black) |
| Monocytes | > 0.7 GIGA/L |
| Basophils | > 0.1 GIGA/L |
| Eosinophils | > 0.5 GIGA/L or<br>> ULN if ULN $\ge 0.5$ GIGA /L |
| Hemoglobin | Males : $\leq 115$ g/L ( $\leq 7.14$ mmol/L), $\geq 185$ g/L ( $11.48$ mmol/L)<br>Females : $\leq 95$ g/L ( $5.9$ mmol/L), $\geq 165$ g/L ( $10.24$ mmol/L)<br>Decrease from Baseline $\geq 20$ g/L ( $1.24$ mmol/L) |
| Hematocrit | Males : $\leq 0.37 \text{ v/v}, \geq 0.55 \text{ v/v}$<br>Females : $\leq 0.32 \text{ v/v}, \geq 0.5 \text{ v/v}$ |
| RBC | ≥ 6 TERA/L |
| Platelets | < 100 GIGA/L |
| Blood pressure | |
| Systolic BP | ≤ 95 mmHg and decrease from baseline ≥ 20 mmHg<br>≥160 mmHg and increase from baseline ≥ 20 mmHg |

Date: 19 AUGUST 2022

Diastolic BP

 $\leq$  45 mmHg and decrease from baseline  $\geq$  10 mmHg  $\geq$ 110 mmHg and increase from baseline  $\geq$  10 mmHg

#### 10.6. Process to Derive Week 48 Data Cut-off

For week 48 evaluations, a strategy for performing the data cut-off for the clinical database was developed, as described in the following:

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

## 10.6.1. Visit Independent Data

Visit independent data (or event-based data) include adverse events, concomitant/prior medication, and surgeries.

## Patients that discontinued study prematurely before or at week 48 (Visit 14)

These patients are defined as having their end of study CRF page filled, and have either:

- a dropout date earlier or equal to date of first injection + 336 days + 5 days (to account for the visit window) or
- a dropout date equal to week 48 visit date

For such patients, all event-based records are kept in the clinical database for week 48 analysis without any change.

## Patients who stayed longer than week 48 (visit 14) in the study

These patients are the patients who did not discontinue study prematurely at/before week 48 (visit 14). Therefore, these patients are either:

- still ongoing after week 48 (visit 14)
- discontinued the study prematurely, but were in the study for longer than week 48 (visit 14)

For such patients, the following will be applied:

All event records with a start date later than the date of the week 48 (visit 14) will be censored. This includes the case where the incomplete date is without any doubt later than the week 48 visit date, eg, week 48 (visit 14) is 10 April 2020 and the incomplete date is May 2020 or only 2021. If the week 48 visit date is missing, then the date of first injection + 336 days will be used instead.

Records with a start date earlier or equal to the date of week 48 (first injection + 336 days if date of week 48 visit is missing) will be kept. This includes records with incomplete dates when the incomplete date is earlier than the week 48 date or in cases where it is not clear if the record occurred before or after week 48 (eg, week 48 [visit 14] is 10 April 2020 and the incomplete date is March 2020, April 2020 or only 2020 or even a missing date). If the date is incomplete, the following adaptions to the data will be made.

#### **Concomitant medication:**

If a stop date is reported which is earlier than the date of week 48 (visit 14) (first injection + 336 days if date of week 48 is missing), the record will not be changed.

If a stop date is reported which is later than the date of week 48 (visit 14) (first injection + 336 days if date of week 48 is missing), the stop date will be set to missing and the variable CMONG will be set to 1 (yes).

## **Adverse Events:**

AEs with a start date on or after the date of the week 48 (visit 14) will be censored. Cut-off date will be first injection + 336 days if date of week 48 is missing.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

If a stop date of adverse event is specified and earlier or equal to date of week 48 (visit 14) (first injection + 336 days if date of week 48 missing), then the record will not be changed.

If a stop date of adverse event is specified and later than the date of week 48 (visit 14) (first injection + 336 days if date of week 48 is missing), then the stop date will be set to missing and the outcome of the adverse event (SAS variable AEOUT) will be set to missing.

If no stop date is specified and the outcome is either not yet reported (AEOUT is blank) or is reported (AEOUT is 3 - recovering/resolving, 4 - not recovered/not resolved, 6 - unknown), then the outcome will be set to missing (AEOUT is blank).

## **Surgeries:**

All surgeries with a date of surgery later than week 48 (visit 14) date will not be included in the analysis. Cut-off date will be first injection + 336 days if date of week 48 is missing.

## **10.6.2.** Study Medication Data

Study medication data in the study eye up to week 44 (visit 13) will be kept for the week 48 analysis. Study medication data in the fellow eye prior to week 48 (week 14) will be included for the week 48 analysis.

## 10.6.3. Visit Dependent Data

All visit dependent data up to week 48 (visit 14) will be kept for the week 48 analysis except for post-dose IOP at the week 48 visit. All visit dependent data later than week 48 (visit 14) will not be included for the week 48 analysis. Unscheduled visits with a date prior to the week 48 (visit 14) visit date will be kept for the week 48 analysis. If a patient did not have a week 48 (visit 14) visit, unscheduled visit will be kept up to date of first injection + 336 days for the week 48 analysis.

#### 10.7. Process to Derive Week 60 Data Cut-off

For week 60 evaluations, the same strategy for performing the data cut-off for the clinical database as described in Appendix 10.6 will be followed. Instead of "first injection + 336 days" for week 48, missing dates for week 60 will be imputed by first injection + 420 days.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

#### 10.8. SAS Procedures

#### 10.8.1. **MMRM**

```
PROC MIXED DATA = <data at Week48>;

CLASS subjid trtpn avisitn basecrt pdme region;

MODEL chg = base basecrt pdme region trtpn avisitn base*avisitn trtpn*avisitn /DDFM=kr;

REPEATED avisitn / SUBJECT=subjid TYPE=un GROUP=trtpn;

LSMESTIMATE trtpn*avisitn "HDq12 - 2q8 " XXX / cl upper testvalue=-4;

*for non-inferiority test with margin = 4;

LSMESTIMATE trtpn*avisitn "HDq16 - 2q8 " XXX / cl upper testvalue=-4;

*for non-inferiority test with margin = 4;

LSMESTIMATE trtpn*avisitn "HDq12 - 2q8 " XXX / cl upper testvalue=0;

*for superiority test;

LSMESTIMATE trtpn*avisitn "HDq16 - 2q8 " XXX / cl upper testvalue=0;

*for superiority test;

RUN;
```

#### **10.8.2. ANCOVA**

```
PROC MIXED DATA = <data until Week48>;

CLASS trtpn basecrt pdme region ;

MODEL chg = base basecrt pdme region trtpn;

LSMESTIMATE trtpn "HDq12 - 2q8" xxx /cl upper testvalue=-4;

*for non-inferiority test with margin = 4;

LSMESTIMATE trtpn "HDq16 - 2q8" xxx /cl upper testvalue=-4;

*for non-inferiority test with margin = 4;

RUN;
```

#### 10.8.3. Multiple Imputation

<u>Step 1. Imputation:</u> Impute missing value using MCMC method and subsequently impute missing data by a regression model.

```
PROC MI DATA=<indata> SEED=01934 OUT=mi01 NIMPUTE=50; * seed = 01934;minimum = 0 0 0 0 0 maximum = 100 100 100 100 100; * BCVA feasible range is 0 to 100; mcmc impute=monotone; VAR base v2 v3 v4 v5;

RUN;

PROC MI DATA=mi01 SEED=01934 out = full NIMPUTE=1; * seed = 01934; minimum = . . . . 0 0 0 0 0 0 maximum = . . . . 100 100 100 100; CLASS basecrt pdme region trtpn

BY _imputation_; MONOTONE REG; VAR basecrt pdme region trtpn base v2 v3 v4 v5;

RUN;
```

## Step 2. Analysis: Each complete dataset is analyzed by ANCOVA model.

```
PROC MIXED DATA = full;

by _imputation_;

CLASS trtpn basecrt pdme region;

MODEL chg = base basecrt pdme region trtpn;

LSMESTIMATE trtpn "HDq12 - 2q8" xxx /cl upper testvalue=-4;

LSMESTIMATE trtpn "HDq16 - 2q8" xxx /cl upper testvalue=-4;

ods output lsmestimates=lsme;

RUN:
```

## **Step 3. Pooling:** The MIANALYZE procedure is used to combine results.

```
PROC MIANALYZE DATA=1sme theta0=-4;

by label;

modeleffects estimate;

stderr stderr;

ods output parameterestimates=parameterest1 VarianceInfo=varinfo1;

run:
```

## 10.8.4. Tipping Point Analysis

Step 1 to Step 3 below are repeated for a range of feasible &delta values. The tipping point will be determined as the &delta value for which the conclusion under MAR is reversed.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

<u>Step 1. Imputation:</u> Impute missing value using MCMC method and subsequently impute missing data by a regression model with MNAR adjustment.

```
PROC MI DATA=<indata> SEED=01934 OUT=mi01 NIMPUTE=50; * seed = 01934; minimum = 0 0 0 0
      maximum = 100 100 100 100 100; * BCVA feasible range is 0 to 100;
      mcmc impute=monotone;
      VAR base v2 v3 v4 v5;
RUN;
PROC MI DATA=mi01 SEED=01934 out = full NIMPUTE=1; * seed = 01934;
      minimum = ...000000
      maximum = . . . . 100 100 100 100 100;
      CLASS basecrt pdme region trtpn
     BY imputation_;
      MONOTONE REG;
      MNAR ADJUST( v5 / SHIFT= &delta ADJUSTOBS=(TRT01PN = 'HDq12') ); * v5 is the outcome at the
visits of interest, e.g. BCVA at week 48;
      MNAR ADJUST( v5 / SHIFT= &delta ADJUSTOBS=(TRT01PN = 'HDq16') );
      VAR basecrt pdme region trtpn base v2 v3 v4 v5;
RUN;
```

# **Step 2. Analysis:** Each complete dataset with MNAR adjustment is analyzed by ANCOVA model.

```
PROC MIXED DATA = full;

by _imputation_;

CLASS trtpn basecrt pdme region;

MODEL chg = base basecrt pdme region trtpn;

LSMESTIMATE trtpn "HDq12 - 2q8" xxx /cl upper testvalue=-4;

LSMESTIMATE trtpn "HDq16 - 2q8" xxx /cl upper testvalue=-4;

ods output lsmestimates=lsme;

RUN;
```

## **Step 3. Pooling:** The MIANALYZE procedure is used to combine results.

Protocol: VGFTe-HD-DME-1934

```
PROC MIANALYZE DATA=1sme theta0=-4;
by label;
modeleffects estimate;
stderr stderr;
ods output parameterestimates=parameterest1 VarianceInfo=varinfo1;
run;
```

## 10.9. Additional Secondary Efficacy Variables and Analyses

This section pre-specifies the statistical approaches for defining and analyzing additional secondary efficacy variables at week 48, for submission to the US FDA (based on the G-SAP that constitutes the primary analysis for the study).

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

## 10.9.1. Analysis Populations

The following populations of analysis will be used for the additional secondary efficacy analyses.

## 10.9.1.1. Full Analysis Set (FAS)

Refer to Section 3.1

#### 10.9.1.2. Modified Full Analysis Set (mFAS)

The modified full analysis set 1 (mFAS1) includes all randomized patients who completed initial treatment phase and maintained their dosing interval (i.e.,

- maintained post 3-dose loading on a q12 interval for HDq12 group and never having their dosing interval shortened to less than q12w;
- maintained post 3-dose loading on a q16 interval for the HDq16 group and never having their dosing interval shortened to less than q16w; and
- all patients in the 2q8 group receive fixed q8 dosing).

The modified full analysis set 2 (mFAS2) includes all randomized patients who completed initial treatment phase and maintained their dosing interval (i.e.,

- maintained post 3-dose loading for All HD group (pooled HDq12 and HDq16 groups) on either q12 or q16 interval and never having their dosing interval shortened to less than q12w; and
- all patients in the 2q8 group receive fixed q8 dosing).

Both analysis sets, mFAS1 and mFAS2, are based on the treatment assigned to the patient at baseline (as randomized).

## 10.9.2. Additional Secondary Efficacy Variable(s)

Additional secondary efficacy analyses will be conducted for the following variables:

- Change from baseline in BCVA (as measured by ETDRS letter score) at week 48 (previously defined primary efficacy variable; see Section 4.5.1)
- Change from 8-weeks post initial treatment phase in BCVA (as measured by ETDRS letter score) at week 48 (additional secondary efficacy variable).

Note that per the dosing schedule shown in Figure 2, the initial treatment phase is through week 8 (3 doses) for both HDq12 and HDq16 treatment groups, and through week 16 (5 doses) for the 2q8 treatment group. Hence 8-weeks post initial treatment phase is Week 16 for both HDq12 and HDq16 treatment groups and Week 24 for the 2q8 treatment group.

## 10.9.3. Additional Secondary Efficacy Analyses

The additional secondary efficacy analyses will be an alternative tipping point analysis on the efficacy variables in Section 10.9.2.

For analysis set (FAS and mFAS) and each variable, the following algorithm will be applied:

1. Within each treatment group, for patients with data at both week 48 and at the designated baseline for the analysis, sort the patient level data for change in BCVA at week 48 from smallest to largest, e.g., ranging from -60, -59, ..., -1, 0, +1, ... to +50 ETDRS letter score. Patients without data at both week 48 and designated baseline are removed from numerator and denominator calculations described below.

Protocol: VGFTe-HD-DME-1934

Date: 19 AUGUST 2022

- 2. For the analysis (sub)set, compare mean change in BCVA at week 48 between HDq12 with the mean change in BCVA at week 48 for the 2q8 control group.
- 3. If the mean change in BCVA for HDq12 group  $\geq$  [mean change in BCVA for 2q8 group  $+ \Delta$ ] where  $\Delta$ =0 or -2, then
  - a. report the number, percentage of patients in the (sub)set relative to the original analysis set, and 2-sided 95% CI (continuity-corrected Wilson (score) method) for HDq12 group,
  - b. report the tipping point value in the HDq12 group analysis subset that is the lowest letter change in BCVA, and
  - c. stop.
- 4. Otherwise, exclude patients with the next worst score in HDq12 group to obtain a new subset. Retain original analysis set in 2q8 control group. Repeat steps 2 and 3, until stopping condition is reached or all patient level data is used in the HDq12 group.

Repeat the above algorithm for HDq16 group and the All HD group.

The above analyses specified for completers may also be repeated using the estimand framework (see Section 5.6).

The reported results from these additional analyses will be as follows (see Table 6).

Table 6: Additional Secondary Efficacy Analyses – Alternative Tipping Point Analyses

| | Population | Variable | Analysis Results | Δ | Tipping<br>Point in<br>HD group |
|---|---|---|---|---|---|
| 1a | FAS <sup>a</sup> | Change from<br>baseline in<br>BCVA at week<br>48 | • Number and Percentage of patients in the HDq12 analysis subset for whom mean change in BCVA ≥ [mean change in BCVA for 2q8 group – Δ] | 0 | x <sub>1</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>HDq16 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | y <sub>1</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>All HD analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | z <sub>1</sub> letters |
| 1b | FASa | Change from<br>baseline in<br>BCVA at week<br>48 | Number and Percentage of patients in the HDq12 analysis subset for whom mean change in BCVA ≥ [mean change in BCVA for 2q8 group − Δ] | -2 | x <sub>2</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>HDq16 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | -2 | y <sub>2</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>All HD analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | -2 | z <sub>2</sub> letters |
| 2a | FASa | Change from<br>8-weeks post<br>initial treatment<br>in BCVA at<br>week 48 | <ul> <li>Number and Percentage of patients in the<br/>HDq12 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | x <sub>3</sub> letters |
| | | WEEK 48 | <ul> <li>Number and Percentage of patients in the<br/>HDq16 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | y <sub>3</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>All HD analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | z <sub>3</sub> letters |

| | Population | Variable | Analysis Results | Δ | Tipping<br>Point in<br>HD group |
|---|---|---|---|---|---|
| 4a | mFAS1 <sup>b</sup> ;<br>mFAS2 <sup>c</sup> | FAS2 <sup>c</sup> 8-weeks post initial treatment in BCVA at | • Number and Percentage of patients in the HDq12 analysis subset for whom mean change in BCVA ≥ [mean change in BCVA for 2q8 group – Δ] | 0 | x <sub>7</sub> letters |
| | week 48 | WEEK 48 | <ul> <li>Number and Percentage of patients in the<br/>HDq16 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | y <sub>7</sub> letters |
| | | | <ul> <li>Number and Percentage of patients in the<br/>All HD analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | 0 | z <sub>7</sub> letters |
| 4b | mFAS1 <sup>b</sup> ; Change from 8-weeks post initial treatment in BCVA at week 48 | <ul> <li>Number and Percentage of patients in the<br/>HDq12 analysis subset for whom mean<br/>change in BCVA ≥ [mean change in<br/>BCVA for 2q8 group – Δ]</li> </ul> | -2 | x <sub>8</sub> letters | |
| | | week 48 | • Number and Percentage of patients in the HDq16 analysis subset for whom mean | -2 | y <sub>8</sub> letters |

Date: 19 AUGUST 2022

change in BCVA ≥ [mean change in

 Number and Percentage of patients in the All HD analysis subset for whom mean change in BCVA ≥ [mean change in

BCVA for 2q8 group  $-\Delta$ ]

BCVA for 2q8 group  $-\Delta$ ]

<sup>&</sup>lt;sup>a</sup> FAS = Full Analysis Set, which includes all randomized patients who received at least 1 dose of study medication.

<sup>&</sup>lt;sup>b</sup> mFAS1 = Modified Full Analysis Set 1, which includes all randomized patients who completed the initial treatment phase and maintained dosing interval (HDq12, HDq16, and 2q8 groups).

<sup>&</sup>lt;sup>c</sup> mFAS2 = Modified Full Analysis Set 2, which includes all randomized patients who completed the initial treatment phase and maintained dosing interval (All HD group and 2q8 group).

## Signature Page for VV-RIM-00208112 v1.0



Signature Page for VV-RIM-00208112 v1.0 Approved